Document: TDOC-0050793 Version: 3.0; Most-Recent; Effective; CURRENT

Status: Effective 



a Novartis company

Name:

Address:

# **Short Title**

# Efficacy and Safety of RTH258 versus Aflibercept

Long Title

# A Two-Year, Randomized, Double-Masked, Multicenter, Three-Arm Study Comparing the Efficacy and Safety of RTH258 versus Aflibercept in Subjects with Neovascular Age-Related Macular Degeneration

| Protocol Number: | RTH258-C001 (formerly TDOC-0016528, Ver | sion 2.0) |
|---|---|---|
| Study Phase: | 3 | |
| Sponsor Name and Address: | Alcon Research, Ltd.<br>6201 South Freeway<br>Fort Worth, Texas 76134-2099 | |
| Investigational Product: | RTH258 solution for intravitreal injection, 6 m mg/50 $\mu L$ | $g/50 \mu L$ and 3 |
| US IND# / EudraCT | IND# 112023 / 2014-004885-95 | |
| Indication Studied: | Neovascular Age-Related Macular Degeneration | on |
| Investigator Agreement: | I have read the clinical study described herein, confidentiality, and agree to conduct the descricompliance with Good Clinical Practices (GCP principles contained within the Declaration of I protocol, and all applicable regulatory requirements. | bed trial in ), the ethical Helsinki, this |
| Principal Investigator: | | |
| | Signature | Date |


Status: Effective 

#### 1 SYNOPSIS

Sponsor: Alcon Research, Ltd. Protocol Number: RTH258-C001

6201 South Freeway Fort Worth, Texas 76134-2099

**Investigational** RTH258, formerly **Study Phase:** 

 $\boxtimes$  3  $\square$  4  $\square$  N/A

Active Ingredient: RTH258

**Protocol Title:** A Two-Year, Randomized, Double-Masked, Multicenter, Three-

Arm Study Comparing the Efficacy and Safety of RTH258 versus Aflibercept in Subjects with Neovascular Age-Related Macular

Degeneration

Investigator(s)/ No. of Sites: Multicenter; Approximately 320 sites

No. of Subjects Duration of Treatment:

Approximately 990 96 weeks

randomized 96 weeks

**Study Population:** Subjects ≥ 50 years of age with untreated active choroidal neovascularization (CNV) secondary to age-related macular degeneration (AMD) in the study eye

**Objective(s):** Primary:

 To demonstrate that RTH258 is not inferior to aflibercept with respect to the change in best-corrected visual acuity (BCVA) from Baseline to Week 48

# Secondary:

- To demonstrate that RTH258 is not inferior to aflibercept with respect to the change in BCVA from Baseline averaged over the period Week 36 to Week 48
- To estimate the proportion of q12 (1 injection every 12 weeks) subjects up to Week 48 in the RTH258 treatment arms
- To estimate the predictive value of the first q12 cycle for maintenance of q12 treatment up to Week 48 in the RTH258 treatment arms
- To evaluate the efficacy of RTH258 relative to aflibercept over the time period up to Week 96 by assessing changes in:

Print Date: Print Date:


Status: Effective 

Sponsor: Alcon Research, Ltd. Protocol Number: RTH258-C001

6201 South Freeway Fort Worth, Texas 76134-2099

o BCVA

- Anatomical parameters of disease activity including central subfield thickness (CSFT) and CNV area
- Presence of 'q8 treatment need' including assessment of q12 status for subjects in the RTH258 3 mg and 6 mg treatment arms
- To assess visual function-related subject-reported outcomes following treatment with RTH258 relative to aflibercept
- To assess the safety and tolerability of RTH258 relative to aflibercept

Methodology:

This study has 3 arms with a 1:1:1 randomization. Subjects in all arms will have visits every 4 weeks through Week 96. The primary analysis will be performed at Week 48.

# Arms 1 and 2 (RTH258):

RTH258 3 mg (Arm 1) and RTH258 6 mg (Arm 2) will be initially injected 3 times at 4 week intervals, at Visit 1/Baseline, Visit 2/Week 4 and Visit 3/Week 8.

Following these loading doses, each subject will be injected every 12 weeks (q12) up to Visit 25/Week 92 unless there is disease activity assessed according to the guidance provided at Visit 6/Week 16, Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 or Visit 22/Week 80. If disease activity is identified, the subject will be reassigned to receive injections every 8 weeks (q8) thereafter, up to study exit. The interactive response technology (IRT) system will make the necessary changes to the dosing per the masked Investigator's assessment. The disease activity assessment will also be performed at Visit 25/Week 92 but will not be entered into IRT and will have no effect on the subject's treatment regimen.

#### Disease Activity Criteria at Week 16:

- Decrease in BCVA of  $\geq 5$  letters compared with Baseline
- Decrease in BCVA of ≥ 3 letters and CSFT increase
   ≥ 75µm compared with Week 12
- Decrease in BCVA of ≥ 5 letters due to neovascular
   AMD disease activity compared with Week 12
- New or worse intraretinal cysts (IRC) / intraretinal fluid (IRF) compared with Week 12

Print Date: Print Date:


Status: Effective 

Sponsor: Alcon Research, Ltd. Protocol Number: RTH258-C001

6201 South Freeway Fort Worth, Texas 76134-2099

#### Disease Activity Criterion at Weeks 20, 32 and 44:

Decrease in BCVA of ≥ 5 letters due to neovascular
 AMD disease activity compared with Week 12

# Disease Activity Criterion at Weeks 56, 68, 80 and 92:

 Decrease in BCVA of ≥ 5 letters due to neovascular AMD disease activity compared with Week 48

# In Arm 3 (aflibercept 2 mg):

2 mg aflibercept, (EYLEA®, comparator) will be injected 3 times at 4 week intervals (Visit 1/Baseline, Visit 2/Week 4 and Visit 3/Week 8), followed by injections q8 up to Visit 25/Week 92.

Treatments: Test Article: RTH258, 3 mg/50 μL and

 $6 \text{ mg}/50 \mu L$ 

**Route of Administration:** Intravitreal (IVT) injection

**Duration of Treatment:** 96 weeks

**Dosage:** 3 mg RTH258 in 50  $\mu$ L (60 mg/mL

formulation)

 $6 \text{ mg RTH}258 \text{ in } 50 \,\mu\text{L} \,(120 \,\text{mg/mL})$ 

formulation)

Control Article: Aflibercept, 2 mg/50 µL

**Route of Administration:** IVT injection

**Duration of Treatment:** 96 weeks

**Dosage:** 2 mg aflibercept in 50 μL

#### Subject Selection: Inclusion Criteria:

- 1. Subjects must give written informed consent before any study related procedures are performed
- 2. Subjects must be 50 years of age or older at Screening
- 3. Active CNV lesions secondary to AMD that affect the central subfield (including retinal angiomatous proliferation [RAP]


Status: Effective 

**Sponsor:** 

Alcon Research, Ltd.
6201 South Freeway
Fort Worth, Texas
76134-2099

lesions with a CNV component) in the study eye, confirmed by the Central Reading Center (CRC) at Screening

- 4. Total area of CNV (including both classic and occult components) must comprise > 50% of the total lesion area in the study eye, confirmed by the CRC at Screening
- 5. Intra and/or subretinal fluid affecting the central subfield of the study eye, confirmed by the CRC at Screening
- 6. BCVA between 78 and 23 letters, inclusive, in the study eye at Screening and Baseline using Early Treatment Diabetic Retinopathy Study (ETDRS) testing

#### **Exclusion Criteria:**

- 1. Any active intraocular or periocular infection or active intraocular inflammation (e.g. infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis) in either eye at Baseline
- 2. Central subfield of the study eye affected by fibrosis or geographic atrophy assessed by color fundus photography and confirmed by the CRC at Screening
- 3. Total area of fibrosis  $\geq$  50% of the total lesion in the study eye, confirmed by the CRC at Screening
- 4. Subretinal blood affecting the foveal center point and/or  $\geq 50\%$  of the lesion of the study eye, confirmed by the CRC at Screening
- 5. Subject has received any approved or investigational treatment for neovascular AMD (other than vitamin supplements) in the study eye at any time
- 6. Any history or evidence of a concurrent intraocular condition in the study eye, including retinal diseases other than neovascular AMD, that, in the judgment of the Investigator, could either require medical or surgical intervention during the course of the study to prevent or treat visual loss that might result from that condition or that limits the potential to gain visual acuity upon treatment with the investigational product
- 7. Retinal pigment epithelium (RPE) rip/tear in the study eye at Screening or Baseline
- 8. Current vitreous hemorrhage or history of vitreous hemorrhage in the study eye within 4 weeks prior to Baseline


Status: Effective 

Sponsor: Alcon Research, Ltd.

6201 South Freeway Fort Worth, Texas 76134-2099

9. History or evidence of the following in the study eye:

• intraocular or refractive surgery within the 90 day period prior to Baseline

Protocol Number: RTH258-C001

- previous penetrating keratoplasty or vitrectomy
- previous panretinal photocoagulation
- previous submacular surgery, other surgical intervention or laser treatment for AMD
- 10. Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 mmHg on medication or according to Investigator's judgment at Screening or Baseline
- 11. Aphakia and/or absence of the posterior capsule in the study eye at Screening or Baseline
- 12. Intra- or periocular use of corticosteroids in the study eye during the 6 month period prior to Baseline
- 13. Use of topical ocular corticosteroids in the study eye for 60 or more consecutive days within the 90 day period prior to Baseline
- 14. Use of systemic corticosteroids for 30 or more consecutive days within the 90 days prior to Baseline, with the exception of low stable doses of corticosteroids (defined as ≤10 mg prednisolone or equivalent dose used for 90 days or more). Inhaled, nasal or dermal steroids are permitted
- 15. Previous therapeutic radiation near the region of the study eye
- 16. Treatment with aflibercept (EYLEA®), bevacizumab (AVASTIN®) or pegaptanib (MACUGEN®) within the 4 week period prior to Baseline, or with ranibizumab (LUCENTIS®) within the 2 week period prior to Baseline in the nonstudy eye
- 17. History of a medical condition (disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding) that, in the judgment of the Investigator, would preclude scheduled study visits, completion of the study, or a safe administration of investigational product
- 18. History of hypersensitivity to any component of the test article, control article, or clinically relevant sensitivity to fluorescein dye (or indocyanine green for subjects in Japan), as assessed by the Investigator
- 19. Pregnant or nursing (lactating) women, where pregnancy is


Status: Effective 

Sponsor: Alcon Research, Ltd.

6201 South Freeway Fort Worth, Texas 76134-2099

defined as the state of a female after conception and until termination of gestation, confirmed by a positive hCG pregnancy test and women of child-bearing potential, defined as all women less than 1 year postmenopausal or less than 6 weeks since sterilization at Baseline, unless they are using effective methods of contraception during dosing of study treatment. Effective contraception methods include:

Protocol Number: RTH258-C001

- Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception
- Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 6 weeks before Baseline. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
- Male sterilization (at least 6 months prior to Baseline). For female subjects in the study, the vasectomized male partner should be the sole partner for that subject
- Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
- Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception
- Placement of an intrauterine device (IUD) or intrauterine system (IUS)
- 20. Participation in an investigational drug, biologic, or device study within 30 days or the duration of 5 half-lives of the investigational product (whichever is longer) prior to Baseline Note: observational clinical studies solely involving over-the-counter vitamins, supplements, or diets are not exclusionary
- 21. Systemic anti-vascular endothelial growth factor (VEGF) therapy within the 90 day period prior to Baseline


Status: Effective 

Sponsor: Alcon Research, Ltd. Protocol Number: RTH258-C001

6201 South Freeway Fort Worth, Texas 76134-2099

22. Stroke or myocardial infarction in the 90 day period prior to Baseline

23. Uncontrolled blood pressure defined as a systolic value  $\geq$  160 mmHg or diastolic value  $\geq$  100 mmHg at Screening

In cases where both eyes are eligible, the eye with the worse BCVA at Baseline will be selected as the study eye. If both eyes have the same BCVA, it is recommended to select the right eye as the study eye.

# Assessments: Efficacy:

- BCVA using ETDRS methodology
- Spectral domain optical coherence tomography (SD-OCT)
- Fluorescein angiography (FA)
- National Eye Institute Visual Function Questionnaire-25 (VFQ-25)

#### Safety:

- General physical exam
- Vital signs
- Blood chemistry/hematology/urinalysis
- Anti-drug antibody (ADA) assessments
- Systemic RTH258 assessments
- Complete ophthalmic exam:
  - o Slit-lamp exam
  - o IOP measurement (pre/postinjection)
  - Fundus exam (dilation at the discretion of the Investigator)
- Postinjection assessments
- Treatment emergent adverse events including events of special interest (ESIs; Section 12.3)

#### Diagnostic:

- Color fundus photography
- Indocyanine green (ICG) imaging (conducted at sites in Japan only)
- Fundus autofluorescence (at a subset of sites)


Status: Effective 

Sponsor: Alcon Research, Ltd. Protocol Number: RTH258-C001

6201 South Freeway Fort Worth, Texas 76134-2099

Endpoints: Primary Efficacy Endpoint:

Change in BCVA from Baseline to Week 48

# **Key Secondary Efficacy Endpoints:**

- Average change in BCVA from Baseline over the period Week 36 through Week 48. For each subject, this endpoint is defined as the average of the changes from Baseline to Weeks 36, 40, 44 and 48
- q12 treatment status at Week 48 (for subjects randomized to RTH258 3 mg and 6 mg only)
- q12 treatment status at Week 48 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg only)

# **Secondary Efficacy Endpoints:**

- Change in BCVA from Baseline to each postbaseline visit
- Average change in BCVA from Baseline over the period Week 84 through Week 96
- Average change in BCVA from Baseline over the period Week 4 to Week 48/96
- Average change in BCVA from Baseline over the period Week 12 to Week 48/96
- Gain in BCVA of 15/10/5 letters or more from Baseline to each postbaseline visit
- Loss in BCVA of 15/10/5 letters or more from baseline to each postbaseline visit
- q12 treatment status at Week 96 (for subjects randomized to RTH258 3 mg and 6 mg)
- q12 treatment status at Week 96 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg)
- Change in CSFT from Baseline to each postbaseline visit
- Change in neurosensory retinal thickness from Baseline to each postbaseline visit
- Change in CNV lesion size from Baseline to Weeks 12, 48 and 96
- Absence of subretinal fluid at each postbaseline visit
- Absence of intraretinal fluid at each postbaseline visit
- Absence of sub RPE fluid at each postbaseline visit
- q8 treatment need status at Weeks 16, 20, 32, 44, 56, 68, 80 and 92

Print Date: Print Date:


Status: Effective 

**Sponsor:** Alcon Research, Ltd.

con Research, Ltd. **Protocol Number: RTH258-C001** 

6201 South Freeway Fort Worth, Texas 76134-2099

> Change in patient reported outcomes (VFQ-25) total and subscale scores from Baseline to Weeks 24, 48, 72 and 96

# Safety Endpoints

- Incidence and characteristics of treatment-emergent adverse events
- Treatment emergent changes in ocular and systemic parameters
- Change in ADAs from Baseline to Weeks 4, 12, 24, 36, 48, 68 and 88
- Extent of systemic RTH258 levels at Weeks 4, 12, 24, 36, 48, 68 and 88

#### **Statistical Methods:**

# Confirmatory testing for efficacy:

**Hypotheses:** The following noninferiority hypotheses are related to a noninferiority margin of 4 letters.

 $_{48}$  = Week 48,  $_{36-48}$  = Week 36 through 48,  $_{R6(3)}$ =RTH258 6(3) mg,  $_{A}$ =Aflibercept 2 mg

**H**<sub>01</sub>:  $\mu_{48R6}$  -  $\mu_{48A} \le$  -4 letters vs **H**<sub>A1</sub>:  $\mu_{48R6}$  -  $\mu_{48A} >$  -4 letters

 $\mathbf{H}_{02}$ : μ<sub>36-48R6</sub> - μ<sub>36-48A</sub>  $\leq$  -4 letters vs  $\mathbf{H}_{A2}$ : μ<sub>36-48R6</sub> - μ<sub>36-48A</sub> > -4 letters

 $\mathbf{H_{03}}$ :  $\mu_{48R3}$  -  $\mu_{48A} \le$  -4 letters vs  $\mathbf{H_{A3}}$ :  $\mu_{48R3}$  -  $\mu_{48A} >$  -4 letters

 $H_{04}$ : μ<sub>36-48R3</sub> - μ<sub>36-48A</sub>  $\leq$  -4 letters vs  $H_{A4}$ : μ<sub>36-48R3</sub> - μ<sub>36-48A</sub> > -4 letters

 $\mu_{48R6}$ ,  $\mu_{48R3}$  and  $\mu_{48A}$  being the corresponding unknown true mean BCVA changes from Baseline to Week 48.

 $\mu_{36\text{-}48R6}$ ,  $\mu_{36\text{-}48R3}$  and  $\mu_{36\text{-}48A}$  are the corresponding unknown true mean values for the average change in BCVA from Baseline over the period Week 36 through 48.

# Primary analysis data set:

The primary efficacy analysis data set is the full analysis set (FAS) with missing values imputed by last observation carried forward (LOCF). The FAS includes all subjects who are randomized and received at least one IVT injection. Sensitivity analyses will be performed using the per protocol analysis set


Status: Effective 

Sponsor: Alcon Research, Ltd. Protocol Number: RTH258-C001

6201 South Freeway Fort Worth, Texas 76134-2099

(PPS) and alternative imputation for missing values including a mixed model repeated measures (MMRM) and observed data only analyses.

# **Statistical testing strategy:**

The 4 hypotheses will be tested in the pre-specified hierarchical sequence according to their numbering (HAn, n=1,2,3,4). Consequently, confirmatory testing of a given hypothesis requires rejection of all preceding null hypotheses. In this setting, each hypothesis will be assessed at a two-sided  $\alpha = 0.05$ , while keeping the global type I error rate at 0.05.

#### Statistical method:

Two-sided 95% confidence intervals (CI) for the differences in means, RTH258 – aflibercept, based on an analysis of variance (ANOVA) model with treatment, Baseline BCVA categories (≤ 55, 56-70, ≥71 letters), and age categories (< 75, ≥ 75 years) as fixed effects will be presented for the primary efficacy analysis. The same ANOVA model will be fitted for the key secondary endpoint, average change in BCVA from Baseline over the period Week 36 through 48.

Within the specified hierarchical testing strategy, noninferiority will be established if the lower limit of the corresponding 95% CI is greater than -4 letters (corresponding to the noninferiority margin of 4 letters).

## Sample size:

A sample size of 297 subjects per treatment arm is sufficient to demonstrate noninferiority (margin = 4 letters) of RTH258 6 mg/3 mg versus aflibercept 2 mg with respect to the BCVA change from Baseline to Week 48 at a two-sided alpha level of 0.05 with a power of approximately 90% assuming equal efficacy and a common standard deviation of 15 letters. A power of at least 90% can be expected for the first key secondary endpoint assuming that averaging over the 4 time points will not lead to an increase in the standard deviation.

To account for a drop-out rate of 10%, a total of 330 subjects will be randomized per treatment arm.


Status: Effective 

#### 1.1 Amendments

#### Amendment 4

Purpose of amendment:

The primary purpose of this amendment is to add back missing text in section 11.3. This text was available in the original protocol, however due to technical issues was accidentally removed and is being added back now. In addition, other minor clarifications have been added to sections 10.5, 10.6, 10.7.4, 12.3.

#### Amendment 3

Purpose of amendment:

The primary purpose of this amendment is to allow ADA analysis of the samples collected from aflibercept treated patients (Section 10.7.5). Minor clarifications have also been made to Sections 9.4, 10.1, 10.9 and 12.3

#### Amendment 2

Note: This TDOC-0050793 was formerly TDOC-0016528, Version 2.0. The change in document numbers was due to a new document management system.

*Purpose of the Amendment:* 

The primary purpose of this amendment is to incorporate changes which resulted from interactions with Regulatory Authorities. In addition, changes have been made to clarify some inclusion/exclusion criteria and study procedures.

Rationale:

**Revision 1** (Section 1. Synopsis, Section 2. Overview of Study Plan, Section 10.2.1. Screening Visit (Day -14 to Day -2) and Section 10.2.2. Visit 1/Baseline (Day 0)): Require BCVA in the study eye to be between 78 and 23 letters, inclusive, at Screening as well as Baseline.

**Rationale:** The purpose of this change is to further clarify the intention of the protocol that the criterion must be met at both the Screening and Baseline Visit by stating it explicitly.

**Revision 2** (Section 1. Synopsis): The term central subfield in exclusion criteria number 4 was changed to foveal center point.


Status: Effective 

**Rationale:** The current wording excludes subjects who are appropriate for anti-VEGF treatment. The change is intended to reduce unnecessary screen failures.

**Revision 3** (Section 1. Synopsis, Section 2. Overview of Study Plan, Section 10.2.2. Visit 1/Baseline (Day 0), Section 10.2.3. Visit 2/Week 4 (Day  $28 \pm 3$  Days) and Visit 3/Week 8 (Day  $56 \pm 3$  Days), Section 10.2.4. Visit 4 (Visit 3 + 1 day) and Section 10.7.5. Analysis of Anti-Drug Antibodies (ADA), Systemic RTH258 and Accumulation (Cmax) of RTH258): Removal of Visit 4 (blood draw for accumulation ( $C_{max}$ ) of RTH258 1 day after the third loading dose) from the protocol.

**Rationale:** This pharmacological assessment will be conducted in another study.

**Revision 4** (Section 2. Overview of Study Plan and Section 10.2.3. Visit 2/Week 4 (Day  $28 \pm 3$  Days) and Visit 3/Week 8 (Day  $56 \pm 3$  Days): Addition of blood draw for ADA and Systemic RTH258 testing to Visit 2/Week 4.

**Rationale:** These tests were added to evaluate the early systemic immune response to the initial intravitreal dose of RTH258 and to determine the systemic exposure of the drug.

**Revision 5** (Section 2. Overview of Study Plan and Section 10.7.16 Postinjection Assessment): Simplification of the postinjection assessment.

**Rationale:** This change is to make post injection fundoscopy at the discretion of the investigator, thereby reducing the risk of postinjection IOP rise due to pupil dilation.

**Revision 6** (Section 10.8. Concomitant Treatment and Section 10.9. Prohibited Treatment): Allowance of all treatments in the nonstudy eye which are approved for exudative AMD in the respective country.

**Rationale:** This change has been made to ensure subjects have unrestricted access to standard of care treatment in the nonstudy eye.

**Revision 7** (Section 13.5. Data Monitoring Committee): Addition of a Data Monitoring Committee (DMC).

**Rationale:** During the Voluntary Harmonization Procedure (VHP) for the RTH258-C002 study, the VHP committee requested that a DMC be established for the C002 study. This DMC will also be utilized to monitor the safety data from study RTH258-C001.

| Alcon - Business Use Only Protocol - Clin Document: TDOC-0050793 Version: 3.0 | nical<br>); Most-Recent; E | Effective Date: 07-Aug-2017 ffective; CURRENT |
|---|---|---|
| Status: Effective | | Page <b>14</b> of <b>8</b> 4 |
| <b>Current Study Status:</b> | | |
| Case Report Form Revision Required: | x Yes | No No |
| Informed Consent Modifications Required: | x Yes | No |
| Applicable Investigators: | x All | Selected (list below) |
| Itemized Changes: | | |
| Notable changes to the protocol are listed in deletions and underlined font for insertions. | - | low using strike through for |
| 1. SYNOPSIS | | |
| Inclusion and Exclusion Criteria | | |
| Inclusion 6 revised: | | |
| BCVA between 78 and 23 letters, inclusive,<br>Early Treatment Diabetic Retinopathy Study | | |
| Exclusion 4 revised: | | |
| Subretinal blood affecting the <u>foveal center</u> of the study eye, confirmed by the CRC at S | _ | field and/or $\geq 50\%$ of the lesion |
| Final paragraph revised: | | |
| In cases where both eyes are eligible, the ey selected as the study eye. If both eyes have right eye as the study eye. | | <u> </u> |
| Assessments | | |
| Removed from Safety: | | |
| Accumulation (Cmax) of RTH258 (in a sub- | set of subjects) | |
| Third and fourth safety endpoints modified: | | |

• Change in ADAs from Baseline to Weeks <u>4</u>, 12, 24, 36, 48, 68 and 88


Status: Effective 

Extent of systemic RTH258 levels at Weeks 8 + 1 day (Cmax) 4, 12, 24, 36, 48, 68 and 88

#### 2. OVERVIEW OF STUDY PLAN

Added to Visit 2/Week 4:

Blood draw for anti-drug antibodies (ADA) and blood draw for systemic RTH258.

Subscript changed:

Visit 4/Visit 3+1 day will be done on a subset of subjects, as determined by IRT, in each treatment arm only applies to a subset of subjects who were randomly selected to complete it and did so before Version 3.0 of the protocol became effective.

Subscript removed:

If BCVA cannot be performed at the Screening Visit, the BCVA may be only performed at the Baseline Visit to qualify the subject.

Subscript changed:

Whether the subject receives an active or sham injection, the study eye will be evaluated 0-5 minutes and 30 (±15) minutes postinjection to ensure that the injection procedure and/or the investigational product have not endangered the health of the eye. This <u>includes an</u> evaluation of central retinal artery perfusion via <u>includes</u> gross assessment of vision status of central retinal artery, presence of retinal detachment, presence of new intraocular hemorrhage(s), and measurement of IOP. <u>Direct visualization to assess the central retinal artery, presence of retinal detachment and presence of new intraocular hemorrhage(s) might be appropriate at the discretion of the investigator and/or based on the results of gross assessment of vision and IOP measurement.</u>

#### 10.2.1. SCREENING VISIT (DAY -14 to DAY -2)

#7 changed:

Perform BCVA on both eyes. If BCVA cannot be performed at the Screening visit the BCVA only performed at the Baseline visit to qualify the subject.


Status: Effective 

# 10.2.2. VISIT 1/BASELINE (DAY 0)

Paragraphs removed/modified:

Subject eligibility will be determined at Screening. However, if the BCVA is not able to be assessed at the Screening Visit, the Baseline Visit BCVA may be used to qualify the subject. Baseline BCVA of the study eye must be between 78 and 23 letters, inclusive, for the subject to qualify.

At the Baseline Visit, subjects will be randomized only if the subject has successfully met all of the eligibility criteria.

At the Baseline Visit IRT will also randomly assign approximately 72 subjects (approximately 24 in each treatment arm; half from Japanese sites and half from non-Japanese sites) to have blood draws for accumulation (Cmax) of RTH258 at Visit 4 (Week 8 + 1 day).

- 12. Contact IRT to obtain a kit number. IRT will also randomly select a subset of subjects to attend Visit 4 (Visit 3+1 day). If the subject is selected for this visit the IRT system will notify the user during this transaction.
- 13. Have the unmasked Investigator perform an IVT injection according to the randomization/kit assignment. The injection procedure may be performed at a later time as long as it occurs within 7 days of the scheduled visit. and within the visit window.

## 10.2.3. VISIT 2/WEEK 4 (DAY 28 ± 3 DAYS) AND VISIT 3/WEEK 8 (DAY 56±3 DAYS)

Added:

- 4. Obtain a blood sample for ADA analysis (Visit 2 only). *Blood draws should take place prior to the IVT injection*.
- 5. Obtain a blood sample for systemic RTH258 analysis (Visit 2 only). *Blood draws should take place prior to the IVT injection.*


Status: Effective 

Changed:

12. 10. Schedule Visit 4 to take place 1 day after Visit 3 if the subject has been predetermined by IRT to attend Visit 4. Otherwise, schedule Visit 5/Week 12 to take place  $84 \pm 7$  days after Visit 1/Baseline.

#### 10.2.4. VISIT 4 (VISIT 3 + 1 DAY)

Changed:

This visit only applies to the subset of subjects who were randomly selected to attend it and did so before Version 3.0 of the protocol became effective.

This visit will be performed on a subset of subjects as determined by IRT.

- 1. Obtain information on any changes in medical health and/or the use of concomitant medications.
- 2. Record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing.
- 3. Obtain a blood sample for C<sub>max</sub> RTH258 analysis.
- 4. Schedule Visit 5/Week 12 to take place 84 ± 7 days after Visit 1/Baseline.

# 10.7.5. ANALYSIS OF ANTI-DRUG ANTIBODIES (ADA), Systemic RTH258 and accumulation (Cmax) of RTH258

Changed:

# 10.7.5. ANALYSIS OF ANTI-DRUG ANTIBODIES (ADA), and Systemic RTH258 and accumulation (Cmax) of RTH258

Collection of blood for ADA; and systemic RTH258, and the accumulation (Cmax) of RTH258 should take place prior to any injection/sham. A standardized procedure for the collection, processing, storage and shipment of these blood samples is provided in a separate laboratory hand book.


Status: Effective 

Only samples from RTH258 treated subjects will be analyzed for ADA, and systemic RTH258. and accumulation (Cmax) of RTH258.

#### 10.7.16. POSTINJECTION ASSESSMENT

First paragraph changed:

The study eye will be assessed before, immediately (0-5 minutes) after and 30 ( $\pm$  15) minutes after each IVT/sham injection to ensure that the procedure and/or the study medication have not endangered the health of the eye. The postinjection assessments include an evaluation of central retinal artery perfusion via a gross assessment of vision (eg, count fingers), the status of the central retinal artery, presence of retinal detachment, presence of new intraocular hemorrhage(s) and measurement of IOP according to the schedule detailed in the MOP. Direct visualization to assess the central retinal artery, presence of retinal detachment, presence of new intraocular hemorrhage(s) might be appropriate at the discretion of the investigator and/or based on the results of gross assessment of vision and IOP measurement.

#### 10.8. Concomitant Treatment

Changed to:

The Investigator should instruct the subject to notify the study site about any new medications he/she takes after enrolling into the study.

Should the nonstudy eye require treatment <u>during the study</u> with an anti-VEGF, <u>ranibizumab</u> a <u>drug which is approved for the treatment of exudative AMD in the respective country</u> should be applied at the discretion of the Investigator and following the procedures established at the respective site. <u>The nonstudy eye treatment may occur at any time once the Baseline study eye injection has been administered.</u>

#### **Table 10-1: Prohibited Treatment**

Nonstudy eye treatment changed to:

Nonstudy eye: <u>Unapproved or Investigational treatment</u> Anti VEGF therapy other than ranibizumab


Status: Effective 

# 13.5. Data Monitoring Committee

Section added:

An independent Data Monitoring Committee (DMC) will be established to monitor the safety of the trial participants, to ensure that the trial is being conducted with the highest scientific and ethical standards, and make appropriate recommendations based on the data seen.

The DMC charter will include the DMC membership and responsibilities, the timing of DMC meetings, the content of the analysis report for the DMC meetings, and the communications with the Sponsor. The DMC will only make recommendations for changes in study conduct.

#### Amendment 1

Purpose of Amendment:

The primary purpose of this amendment is to implement required changes received from regulatory authorities. In addition, the data collection and analysis plan has been changed to improve the reporting of the q12 (treatment every 12 weeks) potential of RTH258 and also clarifications and corrections were implemented based on feedback from key opinion leaders and the CRC.

Rationale:

**Revision 1** (Section 1. Synopsis and Section 11. Analysis Plan): Methodology, endpoints and statistical methods were revised.

**Rationale:** These revisions were made to repeat the analyses performed at Week 48 at the end of the study, and to align with variables measured by the CRC.

**Revision 2** (Section 1. Synopsis): The terms fovea and central fovea in the inclusion and exclusion criteria were changed to central subfield.

**Rationale:** The CRC will use the central subfield for assessing eligibility; this modification was made to provide clarity to Investigators.

**Revision 3** (Section 1. Synopsis): Use of pegaptanib (MACUGEN®) within 4 weeks prior to Baseline added as an excluded medication.

**Rationale:** This addition was made to avoid unnecessary exclusion of subjects with prior exposure to pegaptanib, which is still used in some countries.


Status: Effective 

**Revision 4** (Section 1. Synopsis): Hypersensitivity to povidone iodine was removed as an exclusion.

**Rationale:** Other options are available for preparation of the eye for IVT injection and therefore the original exclusion was unnecessarily restrictive.

**Revision 5** (Section 1. Synopsis): Pregnant and nursing (lactating) women were added to the exclusion criterion.

Rationale: These exclusions were requested by the Japanese Regulatory Authority.

**Revision 6** (Section 1. Synopsis and Section 11.3. Analysis Set): Definition of full analysis set was revised to include all subjects who are randomized and receive at least one IVT injection.

Rationale: This change was requested by the United States Regulatory Agency.

**Revision 7** (Section 2. Overview of Study Plan): Study procedures were revised to state that all blood draws and collection of urine samples should occur prior to subjects receiving an IVT or sham injection or injection of fluorescein dye.

**Rationale:** IVT injection or injection of fluorescein prior to collection of the laboratory samples could confound the results.

**Revision 8** (Section 2. Overview of Study Plan and Section 10.2.5. Visit 5/Week 12 through Visit 25/Week 92): Fluorescein angiography and color fundus photography were added to Visit 5/Week 12.

**Rationale:** An early assessment (Week 12) of fluorescein angiography will allow capture of RTH258 impact on lesion activity compared to aflibercept. Week 12 color fundus photography will allow early assessment of geographic atrophy and identify subjects who have lesions which may have been masked by an increased retinal thickness at Baseline.

**Revision 9** (Section 2. Overview of Study Plan, Figure 10.1.-1: Dosing Schedule by Treatment, Section 10.2.5. Visit 5/Week 12 through Visit 25/Week 92 and Section 10.7.13. Disease Activity Assessment): Disease activity assessment added to Week 92.

**Rationale:** This addition will have no impact on the treatment regimen but will allow the proportion of subjects who can be treated q12 to be estimated at the end of the study (RTH258 3 and 6 mg arms only).


Status: Effective 

**Revision 10** (Section 2. Overview of Study Plan, Section 10.2.2. Visit 1/Baseline, Section 10.2.3. Visit 2/Week 4 and Visit 3/Week 8 and Section 10.2.5. Visit 5/Week 12 through Visit 25/Week 92): Period that the injection may be performed after the scheduled visit was extended from 48 hours to 7 days as long as the injection is performed within the visit window.

**Rationale:** This revision was made to allow more flexibility at the investigative sites while not compromising the study data.

**Revision 11** (Section 10.2.1. Screening Visit): Allowance for screening procedures to be conducted over more than 1 day was added.

**Rationale:** Due to the number and complexity of screening procedures it was determined that it would be beneficial to investigative sites to allow screening to take place over multiple days and will not compromise validity of screening data.

**Revision 12** (Section 10.2.1. Screening Visit): Criteria for rescreening were added.

**Rationale:** These criteria were added to clarify the circumstances under which subjects can be rescreened.

**Revision 13** (Section 10.2.1. Screening Visit): The option for a legally authorized representative to sign the informed consent form was removed.

**Rationale:** This was removed because it was decided that signing of the informed consent form by a legally authorized representative was not appropriate for this trial.

**Revision 14** (Section 10.9. Prohibited Treatment): The allowance for administration of low stable doses of corticosteroids to subjects during the course of the study was added.

Rationale: This was added to clarify and align with the inclusion criteria.

**Revision 15** (Section 11.4.2. Baseline Characteristics): The following baseline characteristics were deleted from the analyses: cyst volume, hyperreflective material, presence of intraocular hemorrhage and central subfield volume.

Rationale: This modification was made to align with the variables captured by the CRC.

**Revision 16** (Section 12.3. Procedures for Recording and Reporting AEs and SAEs): The language regarding adverse events of special interest relative to intraocular inflammation were revised.

| Document: TDOC-0050793 | | | Effective; CURRENT | Date: 07-Aug-2017 |
|---|---|---|---|---|
| Status: Effective | version. | | | Page 22 of 8 |
| <b>Rationale:</b> The grading scales standardization process, and the interest were revised according | erefore the asso | | - | |
| Current Study Status: | | | | |
| Case Report Form Revision Re | equired: | x Yes | No No | |
| Informed Consent Modification | ns Required: | x Yes | No | |
| Applicable Investigators: | | x All | Selecte | ed (list below) |
| Itemized Changes: | | | | |
| Notable changes to the protoco<br>deletions and underlined font for | | he summary b | pelow using strike tl | hrough for |
| 1. SYNOPSIS | | | | |
| Objectives | | | | |
| Objectives revised: | | | | |
| Primary: | | | | |
| <ul> <li>To demonstrate that RT<br/>with respect to the chan<br/>Week 48</li> </ul> | , , | - | | - ' |
| Secondary: | | | | |
| <ul> <li>To demonstrate that RT<br/>with respect to the chan<br/>to Week 48</li> </ul> | , , | | | - ' |
| To estimate the proports | | - | | treatment |
| responders up to Week | | | | 0.10 |
| To estimate the prediction treatment up to Week 4 | | | | <u>of q12</u> |

• To evaluate the efficacy of RTH258 (3mg and 6mg) relative to aflibercept (2mg) over

Printed By: Print Date:

the time period up to Week 96 by assessing changes in:


Status: Effective 

Changes over time in BCVA, central subfield thickness (CSFT) and CNV area

- Absence of any subretinal, intraretinal or sub-retinal pigment epithelium (RPE) fluid-Anatomical parameters of disease activity including central subfield thickness (CSFT) and CNV area
- Presence of 'q8 treatment need' including assessment of q12 status for subjects in the RTH258 3 mg and 6 mg treatment arms disease activity according to protocol defined criteria at Weeks 16, 20, 32, 44, 56, 68 and 80
- To assess visual fundtion-related subject-reported outcomes following treatment with RTH258 relative to aflibercept

# Methodology

Third paragraph of Methodology changed:

Following these loading doses, each subject will be injected every 12 weeks (q12) up to <u>Visit 25/Week 92</u> study exit (Week 96) unless there is the subject meets any of the disease activity assessed according to the guidance provided eriteria at Visit 6/Week 16, Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 or Visit 22/Week 80. If one or more disease activity is identified criteria are met, the subject will be reassigned to receive injections every 8 weeks (q8) thereafter, up to study exit. The interactive response technology (IR) system will make the necessary changes to the dosing per the masked Investigator's assessment. The disease activity assessment will also be performed at Visit 25/Week 92 but will not be entered into IRT and will have no effect on the subject's treatment regimen.

# **Inclusion and Exclusion Criteria**

The following inclusion/exclusion criteria were revised.

Inclusion 3 (this change also applies to inclusion criterion 5 and exclusion criteria 2 and 4): Active CNV lesions secondary to AMD that affect the fovea central subfield (including retinal angiomatous proliferation [RAP] lesions with a CNV component) in the study eye, confirmed by the Central Reading Center (CRC) at Screening

Print Date:


Status: Effective 

Exclusion 16:

Treatment with aflibercept (EYLEA®), or bevacizumab (AVASTIN®) or pegaptanib (MACUGEN®) within the 4 week period prior to Baseline, or with ranibizumab (LUCENTIS®) within the 2 week period prior to Baseline in the nonstudy eye

Exclusion 18:

History of hypersensitivity to any component of the test article, control article, or clinically relevant sensitivity to fluorescein dye or povidone iodine (or indocyanine green for subjects in Japan), as assessed by the Investigator

Exclusion 19:

Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until termination of gestation, confirmed by a positive hCG pregnancy test and Wwomen of child-bearing potential, defined as all women less than 1 year postmenopausal or less than 6 weeks since sterilization at Baseline, unless they are using effective methods of contraception during dosing of study treatment.

# **Endpoints**

Only those with changes are listed.

#### **Key Secondary Efficacy Endpoints:**

- q12 treatment response, defined status at Week 48 (for subjects randomized to RTH258 3 mg and 6 mg only) for a subject in an RTH258 arm who does not meet any disease activity criteria at Week 16 and who, at Week 48, has been maintained on q12 treatment without vision loss (BCVA loss ≤<5 letters at Week 48 compared to Week 12)</li>
- q12 treatment status at Week 48 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg only)

#### **Secondary Efficacy Endpoints:**

- Average change in BCVA from Baseline over the period Week 84 through Week 96
- Average change in BCVA from Baseline over the period Week 4 to Week 48/96
- Average change in BCVA from Baseline over the period Week 12 to Week 48/96


Status: Effective 

q12 treatment status at Week 96 (for subjects randomized to RTH258 3 mg and 6 mg)

- q12 treatment status at Week 96 within the subjects with no q8 need during the first
   q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg)
- Change in neurosensory retinal thickness from Baseline to each postbaseline visit
- Change in area of CNV lesion size from Baseline to Weeks 12, 48 and 96
- Absence of any subretinal, intraretinal or sub RPE fluid at each postbaseline visit
- Absence of intraretinal fluid at each postbaseline visit
- Absence of sub RPE fluid at each postbaseline visit
- Presence of <u>q8</u> treatment need status neovascular AMD disease activity according to protocol defined criteria at Weeks 16, 20, 32, 44, 56, 68, and 80 and 92

## Primary analysis data set

The primary efficacy analysis data set is the full analysis set (FAS) with missing values imputed by last observation carried forward (LOCF). The FAS includes all subjects who are randomized, and received at least one IVT injection. and have a baseline and at least one post baseline measurement of BCVA. Sensitivity analyses will be performed using the per protocol analysis set (PPS) and alternative imputation for missing values including a mixed model repeated measures (MMRM) and analysis of variance (ANOVA) using the FAS with observed data only analyses.

#### 10.1 Outline of Study

Sixth paragraph of Outline of Study was revised:

Following these loading doses, each subject will be injected q12 up to Week 92 study exit (Week 96) unless there is the subject meets any of the disease activity according to the guidance provided eriteria at Visit 6/Week 16, Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 or Visit 22/Week 80. If one or more disease activity criteria are met, disease activity is identified, the subject will be reassigned to receive injections q8 thereafter, up to Week 92 study exit. The IRT system will make the necessary changes to the dosing per the masked Investigator's assessment. The disease activity assessment will also be performed at Visit 25/Week 92 but will not be entered into IRT and will have no effect on the subject's treatment regimen.

Print Date:


Status: Effective 

# 10.2 SCREENING VISIT (DAY -14 TO DAY -2)

Added:

The completion of assessments for this visit may occur on different days. The screening period starts with the first screening procedure (other than signing of the ICF).

One time rescreening of subjects will be allowed in the following circumstances: a) laboratory test(s) need to be repeated, b) when a subject has a temporary medical condition precluding participation. As long as testing can be repeated within 14 days of the first screening, the other screening assessments do not need to be repeated. If rescreening is to occur beyond 14 days from the original screening visit date, then all screening procedures must be repeated. Rescreening will not be permitted for the purpose of capturing new BCVA or imaging assessments that previously failed to qualify the subject. Medical judgment should be exercised to ensure that treatment is not withheld in order for a subject to participate in the study.

#### 10.7.13 DISEASE ACTIVITY ASSESSMENT

Section revised:

The masked Investigator will assess the study eye of all subjects at Visit 6/Week 16, Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 and Visit 22/Week 80. If the subject presents with new or worsening disease activity, as defined in Section 10.1, tThe IRT system will make the necessary changes to the dosing per the masked Investigator's assessment. assign the subject to q8 treatment for the remainder of the study. The disease activity assessment will also be performed at Visit 25/Week 92, but will not be entered into IRT and will have no effect on the subject's treatment regimen. Details of the disease activity assessments are further outlined in the MOP.

#### 11.3 Analysis Sets

Definitions for full analysis set and per protocol analysis set revised:

Full analysis set (FAS): includes all subjects who are randomized, and received at least one IVT injection and have a baseline and at least 1 postbaseline measurement of BCVA. Following the intent-to-treat (ITT) principle, subjects in the FAS will be analyzed according to the treatment group they are assigned at randomization, regardless of whether dosing frequency (q12 to q8) changed at subsequent visits. The FAS will be the primary analysis set for efficacy analyses.


Status: Effective 

The per protocol analysis set (PPS): defined for the primary and key secondary efficacy analysis at Week 48 includes all subjects in the FAS with no protocol deviations that <u>are expected to majorly</u> affect the assessment of efficacy at Week 48 including: lack of compliance (including treatment misallocation), missing data, concomitant medication and deviation from inclusion/exclusion criteria. <u>Discontinuation from treatment due to lack of efficacy does not constitute a reason for exclusion from the PPS.</u>

Before the Week 48 database lock Tthe relevant protocol deviations will be identified specified before the Week 48 database lock in the DEP document and identified at the subject level in the database. Discontinuation from treatment due to lack of efficacy does not constitute a reason for exclusion from the PPS.

#### 11.4.2 BASELINE CHARACTERISTICS

Section revised:

Baseline characteristics will include: primary diagnosis of neovascular AMD, time since diagnosis of neovascular AMD (days), whether neovascular AMD is unilateral or bilateral, BCVA (both as a continuous variable and using categories ( $\leq 55$ , 56-70,  $\geq 71$  letters), lesion type (predominantly classic, minimally classic, pure occult), foveal involvement (subfoveal, extrafoveal, undeterminable), CNV lesion size, presence of sub retinal fluid, presence of intraocular hemorrhage, presence of hyper reflective material, presence of intraretinal fluid/cyst, presence of sub RPE fluid, neurosensory retinal thickness, eyst volume, CSFT (both as a continuous variable and using categories (< 400,  $\ge 400$  µm) and central subfield volume (CSFV).

#### 11.5 Primary and Key Secondary Efficacy Analyses

Only those with changes are listed:

Key Secondary Efficacy Endpoints:

- <u>q12 treatment status at Week 48 (for subjects randomized to RTH258 3 mg and 6 mg only)</u>
- q12 treatment up to Week 48 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg only).
   response, defined for a subject in an RTH258 arm who does not meet any disease activity criteria at Week 16 and who, at Week 48, has been maintained on q12 treatment without vision loss (BCVA loss ≤5 letters at Week 48 compared to Week 12).

Print Date:


Status: Effective 

The primary and key secondary endpoints will be analyzed based on the FAS with last-observation-carried-forward (LOCF) imputation of missing <u>BCVA</u> values (<u>primary and first key secondary endpoint</u>) and a negative q12 treatment status at Week 48 in case of incomplete active treatment up to Week 48 (second and third key secondary endpoint).

#### 11.5.2 STATISTICAL METHODS

Second paragraph was revised:

The proportion of q12 treatment status at Week 48 responders in the RTH258 treatment arms will be presented descriptively together with exact 95% confidence intervals for the proportion of subjects with a positive status: The denominator is all subjects who did not meet disease activity criteria at Week 16, in each RTH258 group. 95% confidence intervals for the observed proportion will also be presented. Subjects who discontinue treatment will be considered as non responders for this analysis.

- For the (overall) proportion of subjects with a positive q12 treatment status at Week 48, the denominator is all FAS subjects in the RTH258 3 mg/6 mg groups, and the numerator is the corresponding number of subjects with no identified q8-need at Week 16, 20, 32 and 44 (while missing the Week 16 assessment is considered as no q8 treatment needed)
- For the predictability of the adequacy of q12 treatment based on the absence of disease activity during the first q12 cycle, the denominator is all FAS subjects in the RTH258 3 mg/6 mg groups with no identified q8-need at Week 16 and Week 20 (while missing the Week 16 assessment is considered a no-q8 treatment needed), and the numerator is the corresponding number of subjects with a positive q12 treatment status at Week 48 ie, with no identified q8-need at Week 16, 20, 32 and 44.

#### 11.5.3 SENSITIVITY ANALYSES

Second paragraph was revised:

Sensitivity analyses to explore the robustness of the primary <u>and first key secondary efficacy</u> <u>analysis results related to missing values will be performed on the observed data in the FAS applying the specified ANOVA model and efficacy analysis results related to missing values will be performed using a mixed model repeated measures (MMRM). Analysis and ANOVA using the FAS with observed data only analyses.</u>

Print Date:


Status: Effective 

#### 11.6 Additional Secondary Efficacy Analyses

Section was revised:

The following secondary efficacy endpoints will be analyzed primarily based on FAS:

- Change in BCVA from Baseline to each postbaseline visit
- Average change in BCVA from Baseline over the period Week 84 through Week 96
- Average change in BCVA from Baseline over the period Week 4 to Week 48/96
- Average change in BCVA from Baseline over the period Week 12 to Week 48/96
- Gain in BCVA of 15/10/5 letters or more from Baseline to each postbaseline visit
- Loss in BCVA of 15/10/5 letters or more from Baseline to each postbaseline visit
- q12 treatment status at Week 96 (for subjects randomized to RTH258 3 mg and 6 mg only)
- q12 treatment status at Week 96 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg only)
- Change in CSFT from Baseline to each postbaseline visit
- Change in neurosensory retinal thickness from Baseline to each postbaseline visit
- Change in area of CNV lesion size from Baseline to Weeks 12, 48 and 96
- Absence of any subretinal, intraretinal or sub RPE fluid at each postbaseline visit
- Absence of intraretinal fluid at each postbaseline visit
- Absence of sub RPE fluid at each postbaseline visit
- Presence of neovascular AMD disease activity according to protocol defined criteria q8-treatment need status assessed at Weeks 16, 20, 32, 44, 56, 68, and 80 and 92
- Change in patient-reported outcomes (VFQ-25) total and subscale scores from Baseline to Weeks 24, 48, 72 and 96

Statistical methods for the analysis of each of the secondary endpoints will be described in the statistical analysis plan (SAP).

#### 11.7 Handling of Missing Data

The primary presentation of efficacy results will use LOCF for the imputation of missing values supplemented by presentations on the observed data only. All non-missing post-baseline values including assessments done at unscheduled visits will be used when implementing the LOCF imputation. <u>Imputations related to the evaluation of the q12-treatment</u> status at Week 96 will follow the concept described for Week 48.


Status: Effective 

# 12.3 Procedures for Recording and Reporting AEs and SAEs

Second and third adverse event of special interest were revised:

• Grade <u>3 aqueous flare and/or Grade 4 aqueous cells</u> <u>4 ocular inflammation</u> (see MOP for grading scale)

• Grade 2 aqueous flare and/or Grade 2 or 3 aqueous cells 2 or 3 ocular inflammation that fails to decrease to 1 or less within 30 days of the onset of the event

Effective Date: 8/7/2017 4:49:40 PM

| | Screening | Visit 1/<br>Baseline | Visit 2/ | Visit 3/ | Visit 47 | Visit 5/ | Visit<br>6/ | Visit 7/ | Visit<br>8/ | Visit 9/ | Visit<br>10/ | Visit<br>11/ | Visit<br>12/ | Visit<br>13/ | Visit<br>14/ |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | Week<br>4 | Week<br>8 | | Week<br>12 | Week<br>16 | Week<br>20 | Week<br>24 | Week<br>28 | Week<br>32 | Week<br>36 | Week<br>40 | Week<br>44 | Week<br>48 |
| | Day<br>-14 to -2 | Day 0 | Day 28 ± 3 Days | Day 56 ± 3 Days | Visit 3<br>+ 1<br>Day | Day<br>84 ± 7<br>Days | Day<br>112 ±<br>7<br>Days | Day<br>140 ±<br>7<br>Days | Day<br>168 ±<br>7<br>Days | Day<br>196 ±<br>7<br>Days | Day 224 ± 7 Days | Day<br>252 ±<br>7<br>Days | Day 280 ± 7 Days | Day<br>308 ±<br>7<br>Days | Day<br>336 ±<br>7<br>Days |
| Informed Consent <sup>1</sup> | X | | | | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | | | |
| Medical History/<br>Concomitant<br>Medications | X | | | | | | | | | | | | | | |
| Changes in<br>Concomitant<br>Medications | | X | X | X | | X | X | X | X | X | X | X | X | X | X |
| Monitor for Adverse<br>Events | X | X | X | X | | X | X | X | X | X | X | X | X | X | X |
| Inclusion/ Exclusion | X | $X^2$ | | | | | | | | | | | | | |
| Visual Function<br>Questionnaire-25<br>(VFQ-25) <sup>3</sup> | | X | | | | | | | X | | | | | | X |
| General Physical<br>Exam <sup>4</sup> | X | | | | | | | | | | | | | | X |
| Vital Signs | X | X | X | X | | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Test <sup>5</sup> | X | | | | | | | | | | | | | | X |
| Blood/Urine<br>Sample: Chemistry/<br>Hematology/<br>Urinalysis <sup>6</sup> | X | | | | | X | | | | | | | | | X |
| Blood Draw for<br>Anti-Drug<br>Antibodies (ADA) <sup>6</sup> | | X | X | | | X | | | X | | | X | | | X |
| Blood Draw for<br>Systemic RTH258 <sup>6</sup> | | X | X | | | X | | | X | | | X | | | X |
| Best-Corrected<br>Visual Acuity<br>(BCVA) | $X^8$ | $X^8$ | X | X | | X <sup>8</sup> | X | X | X <sup>8</sup> | X | X | X <sup>8</sup> | X | X | X <sup>8</sup> |
| Complete Ophthalmic Exam <sup>9</sup> | X <sup>8</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | $X^8$ |

Printed By:

2

**OVERVIEW OF STUDY PLAN** 

| Status: Effective | Document: TDOC-0050793 | Alcon - Business Use Only Protocol - Clinical |
|---|---|---|
| | Version: 3.0; Most-Recent; Effective; CURRENT | Protocol - Clinical |
| | Effective; | |
| | CURRENT | Effective |

| | Day<br>-14 to -2 | Visit 1/<br>Baseline<br>Day 0 | Visit 2/ Week 4 Day 28 ± 3 Days | Visit 3/ Week 8 Day 56 ± 3 Days | Visit 4 <sup>7</sup> Visit 3 + 1 Day | Visit 5/ Week 12 Day 84 ± 7 Days | Visit 6/ Week 16 Day 112 ± 7 Days | Visit 7/ Week 20 Day 140 ± 7 Days | Visit 8/ Week 24 Day 168 ± 7 Days | Visit 9/ Week 28 Day 196 ± 7 Days | Visit 10/ Week 32 Day 224 ± 7 Days | Visit 11/ Week 36 Day 252 ± 7 Days | Visit 12/ Week 40 Day 280 ± 7 Days | Visit 13/ Week 44 Day 308 ± 7 Days | Visit 14/ Week 48 Day 336 ± 7 Days |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Spectral Domain<br>Optical Coherence<br>Tomography (SD-<br>OCT) | X <sup>8</sup> | X | X | X | | X | X | X | X | X | X | X | X | X | X <sup>8</sup> |
| Fluorescein<br>Angiography (FA) <sup>10</sup> | $X^8$ | | | | | X | | | | | | | | | $X^8$ |
| Color Fundus<br>Photography | X <sup>8</sup> | | | | | X | | | | | | | | | X <sup>8</sup> |
| Indocyanine Green (ICG) <sup>11</sup> | X <sup>8</sup> | | | | | | | | | | | | | | |
| Fundus Autofluorescence (FAF) <sup>12</sup> | | X <sup>12</sup> | | | | X <sup>12</sup> | | | | | | | | | $X^{12}$ |
| Disease Activity Assessment | | | | | | | X | X | | | X | | | X | |
| Contact Interactive<br>Response<br>Technology (IRT) | X | X | X | X | | | X | X | X | X | X | X | X | X | X |
| Administer Study<br>Injection or Sham <sup>13</sup> /<br>Postinjection<br>Assessment <sup>14</sup> | | X | X | X | | | X | X | X | X | X | X | X | X | X |

| Status: Effective | Document: TDOC-0050793 | Alcon - Business Use Only Protocol - Clinical |
|---|---|---|
| | Version: 3.0; Most-Recent; Effective; CURRENT | rotocol - Clinical |
| | Effective; | |
| | ; CURRENT | Effective Date: 8/7/2017 4:49:40 |

| | Visit<br>15/<br>Week<br>52 | Visit<br>16/<br>Week<br>56 | Visit<br>17/<br>Week<br>60 | Visit<br>18/<br>Week<br>64 | Visit<br>19/<br>Week<br>68 | Visit<br>20/<br>Week<br>72 | Visit<br>21/<br>Week<br>76 | Visit<br>22/<br>Week<br>80 | Visit<br>23/<br>Week<br>84 | Visit<br>24/<br>Week<br>88 | Visit<br>25/<br>Week<br>92 | Visit 26/<br>Week 96 /<br>Exit 15 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day<br>364 ±<br>7<br>Days | Day<br>392 ±<br>7<br>Days | Day<br>420 ±<br>7<br>Days | Day<br>448 ±<br>7<br>Days | Day<br>476 ±<br>7<br>Days | Day<br>504 ±<br>7<br>Days | Day 532 ± 7 Days | Day<br>560 ±<br>7<br>Days | Day<br>588 ±<br>7<br>Days | Day<br>616 ±<br>7<br>Days | Day<br>644 ±<br>7<br>Days | Day<br>672 ±<br>7<br>Days |
| Changes in Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Monitor for Adverse<br>Events | X | X | X | X | X | X | X | X | X | X | X | X |
| Visual Function<br>Questionnaire-25 (VFQ-25) <sup>3</sup> | | | | | | X | | | | | | X |
| General Physical Exam <sup>4</sup> | | | | | | | | | | | | X |
| Vital Signs | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy<br>Test <sup>5</sup> | | | | | | | | | | | | X |
| Blood/Urine Sample:<br>Chemistry/ Hematology/<br>Urinalysis <sup>6</sup> | | | | | | | | | | | | X |
| Blood Draw for Anti-Drug<br>Antibodies (ADA) <sup>6</sup> | | | | | X | | | | | X | | $(X)^{16}$ |
| Blood Draw for Systemic<br>RTH258 <sup>6</sup> | | | | | X | | | | | X | | $(X)^{16}$ |
| Best-Corrected Visual<br>Acuity (BCVA) | X | X | X <sup>8</sup> | X | X | X <sup>8</sup> | X | X | X <sup>8</sup> | X | X | X <sup>8</sup> |
| Complete Ophthalmic<br>Exam <sup>9</sup> | X | X | X | X | X | X | X | X | X | X | X | $X^8$ |
| Spectral Domain Optical<br>Coherence Tomography<br>(SD-OCT) | X | X | X | X | X | X | X | X | X | X | X | $X^8$ |
| Fluorescein Angiography (FA) <sup>10</sup> | | | | | | | | | | | | $X^8$ |
| Color Fundus Photography | | | | | | | | | | _ | _ | $X^8$ |
| Fundus Autofluorescence (FAF) <sup>12</sup> | | | | | | | | | | | | X <sup>12</sup> |

| | Visit<br>15/<br>Week<br>52 | Visit<br>16/<br>Week<br>56 | Visit<br>17/<br>Week<br>60 | Visit<br>18/<br>Week<br>64 | Visit<br>19/<br>Week<br>68 | Visit<br>20/<br>Week<br>72 | Visit<br>21/<br>Week<br>76 | Visit<br>22/<br>Week<br>80 | Visit<br>23/<br>Week<br>84 | Visit<br>24/<br>Week<br>88 | Visit<br>25/<br>Week<br>92 | Visit 26/<br>Week 96 /<br>Exit <sup>15</sup> |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Day<br>364 ±<br>7<br>Days | Day<br>392 ±<br>7<br>Days | Day<br>420 ±<br>7<br>Days | Day<br>448 ±<br>7<br>Days | Day<br>476 ±<br>7<br>Days | Day<br>504 ±<br>7<br>Days | Day<br>532 ±<br>7<br>Days | Day<br>560 ±<br>7<br>Days | Day<br>588 ±<br>7<br>Days | Day<br>616 ±<br>7<br>Days | Day<br>644 ±<br>7<br>Days | Day<br>672 ±<br>7<br>Days |
| Disease Activity Assessment | | X | | | X | | | X | | | X | |
| Contact Interactive<br>Response Technology<br>(IRT) | X | X | X | X | X | X | X | X | X | X | X | |
| Administer Study<br>Injection or Sham <sup>13</sup> /<br>Postinjection Assessment <sup>14</sup> | X | X | X | X | X | X | X | X | X | X | X | |
| Complete Exit Form <sup>15</sup> | | | | | | | | | | | | X |

- 1. The informed consent form must be signed/dated prior to performing any study procedures, including screening procedures.
- 2. Verify that inclusion/exclusion criteria are met at Visit 1/Baseline prior to assignment of study treatment.
- 3. Questionnaires are to be administered at those sites where validated translations are available and where they are approved by the corresponding Independent Ethics Committee/Institutional Review Board (IEC/IRB). Questionnaires must be administered prior to any examination.
- 4. All clinically significant findings will be recorded as medical history or adverse events, as appropriate.
- 5. Required for all female subjects of childbearing potential. Urine pregnancy tests will be performed unless local regulations require a serum pregnancy test.
- 6. All blood draws and urine collections should be performed prior to receiving the IVT or sham injection and prior to injection of fluorescein dye.
- 7. Visit 4/Visit 3+1 day only applies to the subset of subjects who were randomly selected to complete it and did so before Version 3.0 of the protocol became effective.
- 8. Both eyes; all other assessments are study eye only.
- 9. Includes slit-lamp exam, IOP measurement, and fundus exam. Dilation for the fundus exam is at the discretion of the Investigator.
- 10. Other FA assessments, done outside of the visit schedule, may be performed at Investigator's discretion based on exam findings, observations, etc.
- 11. ICG imaging applies to subjects screened at sites in Japan only.
- 12. FAF will be performed at a subset of sites.
- 13. Subjects will be randomized to one of the following treatments: RTH258 3 mg, RTH258 6 mg, or aflibercept 2 mg. Beginning at Week 16, when subjects do not receive an active injection, they will receive a sham injection. The injection may be performed at a later time, as long as it is within 7 days of the scheduled visit and within the visit window.
- 14. Whether the subject receives an active or sham injection, the study eye will be evaluated 0-5 minutes and 30 (±15) minutes postinjection to ensure that the injection procedure and/or the investigational product have not endangered the health of the eye. This includes an evaluation of central retinal artery perfusion via gross assessment of vision and measurement of IOP. Direct visualization to assess the central retinal artery, presence of retinal detachment and presence of new

intraocular hemorrhage(s) might be appropriate at the discretion of the investigator and/or based on the results of gross assessment of vision and IOP measurement.

- 15. All exit procedures should be followed, regardless of when the subject exits the study.
- 16. Blood draws for ADA and systemic RTH258 will be performed if the subject exits at or before Visit 24/Week 88.

Alcon - Business Use Only Protocol - Document: TDOC-0050793 Version Status: Effective

Version: 3.0; Most-Recent; Effective; CURRENT


Status: Effective 

# 3 ABBREVIATIONS

| Abbreviation | Definition |
|--------------|--------------------------------------------|
| ADA | Anti-drug antibody |
| AE | Adverse event |
| AEF | Adverse event form |
| AMD | Age-related macular degeneration |
| ANOVA | Analysis of variance |
| BCVA | Best-corrected visual acuity |
| CI | Confidence interval |
| CNV | Choroidal neovascularization |
| CRC | Central reading center |
| CRF | Case report form |
| CSFT | Central subfield thickness |
| CSM | Clinical site management |
| CTM | Clinical trial management |
| DEP | Deviations and evaluability plan |
| DMC | Data Monitoring Committee |
| EDC | Electronic data capture |
| ESI | Event of special interest |
| ETDRS | Early treatment diabetic retinopathy study |
| FA | Fluorescein angiography |
| FAF | Fundus autofluorescence |
| FAS | Full analysis set |
| GCP | Good clinical practice |
| ICF | Informed consent form |
| ICG | Indocyanine green |
| ICH | International Conference on Harmonization |
| IEC | Independent ethics committee |
| IOP | Intraocular pressure |
| IP | Investigational product |
| IRB | Institutional review board |
| IRC | Intraretinal cysts |
| IRF | Intraretinal fluid |
| IRT | Interactive response technology |
| ITT | Intent-to-treat |
| IUD | Intrauterine device |
| IUS | Intrauterine system |
| IVT | Intravitreal |
| LOCF | Last observation carried forward |
| mg | Miligram |
| mL | Milliliter |
| mmHg | Millimeters of mercury |
| MMRM | Mixed model repeated measures |
| MOP | Manual of procedures |

Status: Effective 

| Abbreviation | Definition |
|--------------|-----------------------------------------------|
| PCV | Polypoidal choroidal vasculopathy |
| PPS | Per protocol analysis set |
| PRN | Pro re nata |
| q8 | Every 8 weeks |
| q12 | Every 12 weeks |
| RAP | Retinal angiomatous proliferation |
| RPE | Retinal pigment epithelium |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| scFv | Single chain variable fragment |
| SD-OCT | Spectral-domain optical coherence tomography |
| SUSAR | Suspected unexpected serious adverse reaction |
| μL | Microliter |
| VEGF | Vascular endothelial growth factor |
| VFQ-25 | Visual Function Questionnaire |
| VHP | Voluntary Harmonization Process |

## **Glossary of Terms**

| Term | Definition |
|---|---|
| AMD | Clinical and/or angiographic signs of retinal degeneration (including drusen, |
| | hypo- or hyper-pigmentation, geographic atrophy, and choroidal |
| | neovascularization) with no other likely etiologic explanations for the |
| | degenerative changes |
| Central | The circular area within 1 mm diameter around the foveal center on imaging |
| Subfield | |
| CNV | Angiographic evidence of new blood vessel growth within the central |
| (subfoveal) | subfield. The lesion containing the new vessel growth may be classic and/or |
| secondary to | occult and can include thick contiguous blood or an area of elevated blocked |
| AMD | fluorescence corresponding to pigment that obscures the boundaries of the |
| | neovascular components, or serous detachment of the retinal pigment |
| | epithelium |

 ${\bf Alcon \textbf{-} Business} \ Use \ Only \ {\tt Protocol} \ \textbf{-} \ {\tt Clinical}$ 

Document: TDOC-0050793

Version: 3.0; Most-Recent; Effective; CURRENT

Effective Date: 07-Aug-2017

Status: Effective 

| 4 | $T_{\Lambda}$ | RI. | $\mathbf{F}$ | $\mathbf{OF}$ | CO | N | ΓEN | T | C |
|---|---|---|---|---|---|---|---|---|---|
| T | | | | $O_{\mathbf{I}}$ | $\mathbf{v}$ | T 4 1 | | | J |

| 1 | SYNOPSIS | 2 |
|---|---|---|
| 1.1 | Amendments | 12 |
| 2 | OVERVIEW OF STUDY PLAN | 31 |
| 3 | ABBREVIATIONS | 36 |
| 4 | TABLE OF CONTENTS | 38 |
| List of Ta | bles | 40 |
| List of Fig | gures | 40 |
| 5 | INTRODUCTION | 41 |
| 5.1 | Study Rationale and Background | 41 |
| 5.1.1 | Dose Rationale | 43 |
| 5.1.2 | Treatment Regimen Rationale | 43 |
| 5.2 | Benefits and Potential Risks | 44 |
| 6 | ETHICS | 45 |
| 7 | PROTOCOL AMENDMENTS | 46 |
| 8 | SUBJECT POPULATION | 46 |
| 9 | TREATMENTS ADMINISTERED | 46 |
| 9.1 | Identity of Study Treatments | 46 |
| 9.2 | Usage | 47 |
| 9.3 | Accountability Procedures | 48 |
| 9.4 | Subject Confidentiality and Methods Used to Minimize Bias | 48 |
| 10 | STUDY PROCEDURES | 50 |
| 10.1 | Outline of Study | 50 |
| 10.2 | Visits and Examinations | 52 |
| 10.2.1 | Screening Visit (Day -14 to Day -2) | 52 |
| 10.2.2 | Visit 1/Baseline (Day 0) | |
| 10.2.3 | Visit 2/Week 4 (Day $28 \pm 3$ Days) and Visit 3/Week 8 (Day $56 \pm 3$ Days) | 55 |
| 10.2.4 | Visit 4 (Visit 3 + 1 Day) | 56 |
| 10.2.5 | Visit 5 /Week 12 (Day 84 ± 7 Days) Through Visit 25 /Week 92 (Day 64-7 Days) | |
| 10.2.6 | Visit 26/Week 96/Exit Visit (Day 672 ± 7 Days) or Early Exit | |
| 10.3 | Unscheduled Visits | |

| | TDOC-0050793 Version: 3.0; Most-Recent; Effective; CURRE | ve Date: 07-Aug-2017<br>NT<br>Page <b>39</b> of <b>84</b> |
|---|---|---|
| 10.4 | Discontinued Subjects | C |
| 10.5 | · · | |
| | Discontinuation of Study Treatment | |
| 10.6 | Clinical Study Termination | |
| 10.7 | Study Methods and Measurements | 61 |
| 10.7.1 | Visual Function Questionnaire-25 | 61 |
| 10.7.2 | General Physical Exam and Vital Signs | 61 |
| 10.7.3 | Pregnancy Test | 61 |
| 10.7.4 | Laboratory Analysis of Blood and Urine | 62 |
| 10.7.5 | Analysis of Anti-drug Antibodies (ADA) and Systemic RT | H25862 |
| 10.7.6 | Best-Corrected Visual Acuity | 62 |
| 10.7.7 | Complete Ophthalmic Examination | 62 |
| 10.7.8 | Spectral Domain Optical Coherence Tomography Imaging | |
| 10.7.9 | Fluorescein Angiography | |
| 10.7.10 | Color Fundus Photography | |
| 10.7.11 | Indocyanine Green | |
| 10.7.12 | Fundus Autofluorescence | |
| 10.7.13 | Disease Activity Assessment | |
| 10.7.14 | Intravitreal Administration of Investigational Product | |
| 10.7.15 | Administration of Sham Injection | |
| 10.7.16 | Postinjection Assessment | |
| 10.8 | Concomitant Treatment | 65 |
| 10.9 | Prohibited Treatment | 65 |
| 11 | ANALYSIS PLAN | 66 |
| 11.1 | General Considerations | 66 |
| 11.2 | Subject Evaluability | 66 |
| 11.3 | Analysis Sets | 66 |
| 11.4 | Demographic and Baseline Characteristics | 67 |
| 11.4.1 | Demographic Characteristics | 67 |
| 11.4.2 | Baseline Characteristics | 67 |
| 11.5 | Primary and Key Secondary Efficacy Analyses | 68 |
| 11.5.1 | Statistical Hypotheses | 68 |
| 11.5.2 | Statistical Methods | 69 |
| 11.5.3 | Sensitivity Analyses | 70 |
| 11.5.4 | Subgroups | 70 |
| 11.6 | Additional Secondary Efficacy Analyses | 70 |
| 11.7 | Handling of Missing Data | 71 |

| | usiness Use Only Protocol - Clinical Effective Date TDOC-0050793 Version: 3.0; Most-Recent; Effective; CURRENT | e: 07-Aug-2017 |
|---|---|---|
| Status: Effe | | Page <b>40</b> of <b>84</b> |
| 11.8 | Multiplicity | 71 |
| 11.9 | Safety | 72 |
| 11.9.1 | Treatment Exposure | 72 |
| 11.9.2 | Medical History | 72 |
| 11.9.3 | Concomitant Therapies | 72 |
| 11.9.4 | Safety Parameters | 72 |
| 11.9.5 | Adverse Events | 73 |
| 11.10 | Interim Analyses | 73 |
| 11.11 | Sample Size Justification | 73 |
| 12 | ADVERSE EVENTS | 74 |
| 12.1 | General Information | 74 |
| 12.2 | Monitoring for Adverse Events | 74 |
| 12.3 | Procedures for Recording and Reporting AEs and SAEs | 75 |
| 12.4 | Intensity and Causality Assessments | 78 |
| 12.5 | Unmasking of the Study Treatment | 79 |
| 12.6 | Follow-Up of Subjects with Adverse Events | 79 |
| 12.7 | Pregnancy in the Clinical Trial | 79 |
| 13 | DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS | 80 |
| 13.1 | Completion of Source Documents and Electronic Case Report Form | ns80 |
| 13.2 | Data Review and Clarifications | 81 |
| 13.3 | Regulatory Documentation and Records Retention | 81 |
| 13.4 | Quality Assurance and Quality Control | 81 |
| 13.5 | Data Monitoring Committee | 82 |
| 14 | REFERENCES | 82 |
| 15 | APPENDIX | 84 |
| | List of Tables | |
| Table 10-1 | Prohibited Medication | 66 |
| | List of Figures | |
| Figure 10- | 1 Dosing Schedule by Treatment | 52 |


Status: Effective 

#### 5 INTRODUCTION

## 5.1 Study Rationale and Background

Age-related macular degeneration (AMD) is the leading cause of severe vision loss in people affecting 10%-13% of individuals over the age of 65 in North America, Europe, and Australia (Kawasaki 2010, Rein 2009, Smith 2001). Genetic, environmental and health factors play an important role in the pathogenesis of the disease.

AMD is classified into 2 clinical subtypes: the non-neovascular (atrophic) or dry form and the neovascular (exudative) or wet form (Ferris 1984, Lim 2012, Miller 2013). Neovascular AMD is characterized by the growth of abnormal new blood vessels (neovascularization) under the retinal pigment epithelium (RPE) or subretinal space from the subjacent choroid, termed choroidal neovascularization (CNV) (Ferris, 1984). These newly formed vessels have an increased likelihood to leak blood and serum, damaging the retina by stimulating inflammation and scar tissue formation. This damage to the retina results in progressive, severe, and irreversible vision loss (Shah 2007, Shah 2009). Without treatment, most affected eyes will have poor central vision (20/200) within 12 months (TAP 2003). Although the neovascular form of the disease is only present in about 10% of all AMD cases, it accounted for approximately 90% of the severe vision loss from AMD prior to the introduction of antivascular endothelial growth factor (VEGF) treatments (Ferris 1983, Sommer 1991, Wong 2008).

VEGF has been shown to be elevated in patients with neovascular AMD and is thought to play a key role in the neovascularization process (Spilsbury 2000). The use of intravitreal (IVT) pharmacotherapy targeting VEGF has significantly improved visual outcomes in patients with neovascular AMD (Bloch 2012, Campbell 2012). Anti-VEGF treatments, such as ranibizumab (LUCENTIS®) and aflibercept (EYLEA®), inhibit VEGF signaling pathways and have been shown to halt the growth of neovascular lesions and resolve retinal edema.

#### **Ranibizumab**

In two Phase 3 studies of ranibizumab with monthly dosing regimens, approximately 95% of ranibizumab treated subjects experienced stabilization of vision (defined as a loss of fewer than 15 early treatment diabetic retinopathy study [ETDRS] letters) or improvement in vision at 12 months compared with 62% and 64% in the control groups (Rosenfeld 2006, Brown 2009). Twenty-five to 40% of subjects in the ranibizumab groups gained  $\geq$  15 letters at 12 months compared with 5-6% in the 2 control groups. On average, ranibizumab treated


Status: Effective 

subjects gained 7-11 letters of vision after 12 months, whereas control subjects lost an average of approximately 10 letters. This gain in visual acuity was essentially maintained during the second year of both Phase 3 studies while vision, on average, continued to decline in the control group. The visual acuity benefits, which indicate a suspension of neovascular AMD rather than a slowdown of its progression, were supported by corresponding effects on lesion anatomy and subject reported outcomes. The latter demonstrated statistically and clinically meaningful improvements in near activities, distance activities, and vision specific dependency as measured by the National Eye Institute Visual Function Questionnaire-25 (VFQ-25).

#### **Aflibercept**

In two parallel Phase 3 trials of aflibercept, treatment naïve subjects with neovascular AMD were randomized to 2 doses (0.5 and 2.0 mg) and 2 regimens (every 4 weeks and every 8 weeks with 2.0 mg) or the control arm (ranibizumab 0.5 mg every 4 weeks). At 52 weeks, all aflibercept groups, independent of doses and regimens, were noninferior to the ranibizumab group with equal stabilization of vision in 95% of eyes (Heier 2012). In the 2 mg aflibercept every 4 weeks group, there was a mean best-corrected visual acuity (BCVA) improvement of 9.3 letters and in the 2 mg aflibercept every 8 weeks group there was an improvement of 8.4 letters compared to the control group which had a mean improvement of 8.7 letters. In the second year of the study subjects were switched to a capped (treatment required at least every 12 weeks) pro re nata (PRN) regimen. The proportion of subjects who maintained BCVA ranged between 91% and 92% for all groups. Mean BCVA improvements ranged from 7.9 (ranibizumab), 7.6 (aflibercept 2 mg every 4 weeks and every 8 weeks) to 6.6 (aflibercept 0.5 mg every 4 weeks). The retreatment frequency was similar between the aflibercept and ranibizumab arms during the capped PRN year, with a mean of 4.1 injections for the aflibercept 2 mg every 4 weeks arm, 4.2 injections for the aflibercept 2 mg every 8 weeks arm and 4.7 for the ranibizumab arm (Schmidt-Erfurth 2014).

#### **RTH258**

RTH258, formerly known as ESBA1008, is a humanized single-chain Fv (scFv) antibody fragment inhibitor of VEGF with a molecular weight of ~26 kDa that is being developed for the treatment of CNV associated with neovascular AMD. It is an inhibitor of VEGF-A and works by binding to the receptor binding site of the VEGF-A molecule, thereby preventing the interaction of VEGF-A with its receptors VEGFR1 and VEGFR2 on the surface of endothelial cells. Increased levels of signaling through the VEGF pathway are associated with pathologic ocular angiogenesis and retinal edema. Inhibition of the VEGF pathway has


Status: Effective 

been shown to inhibit the growth of neovascular lesions and resolve retinal edema in patients with neovascular AMD.

In an ascending single dose study, Alcon protocol C-10-083, several doses of RTH258 (0.5, 3.0, 4.5 and 6 mg), were evaluated versus ranibizumab 0.5 mg with regard to the mean change from Baseline to Month 1 in central subfield thickness (CSFT) as measured by spectral-domain optical coherence tomography (SD-OCT) (primary efficacy endpoint). Treatment with RTH258 provided similar reductions for all doses in CSFT to ranibizumab. The primary statistical analysis compared RTH258 4.5 mg and 6.0 mg versus ranibizumab 0.5 mg with both doses achieving noninferiority. Notable however was the median time to receiving standard of care which was longer for the RTH258 3.0 mg, 4.5 mg and 6.0 mg doses (75 days in the 6.0 mg group compared with 45 days in the ranibizumab group), suggesting a longer duration of treatment effect. RTH258 6 mg was the highest dose tested in the study and no unexpected safety issues were reported that would preclude further clinical development.

Subsequently the safety and efficacy of the RTH258 6 mg dose were evaluated versus aflibercept 2 mg in a 56 week multiple dose study (Alcon protocol C-12-006) with a primary endpoint at 12 weeks. The efficacy data from this study showed that RTH258, when it was given every 8 weeks (q8), was as effective as the active control in terms of BCVA change from Baseline. There were numerical advantages with RTH258 over aflibercept with regard to the change in CSFT from Baseline. The majority (72%) of the RTH258 treated subjects who completed an extension of the study, who received treatment every 12 weeks (q12), showed visual stability. There were no adverse events in the RTH258 group that negatively differentiated the drug from the control. The majority of adverse events were mild or moderate in nature and either resolved spontaneously or with treatment.

#### **5.1.1 Dose Rationale**

C-10-083 and C-12-006 suggest that a 6 mg dose of RTH258 is effective and safe. The RTH258 3 mg dose is included in order to evaluate the dose-response relationship following multiple dosing with RTH258.

# **5.1.2** Treatment Regimen Rationale

While VEGF inhibitors have vastly improved patient outcomes for neovascular AMD, there still remains a need for treatments and regimens which offer a reduced frequency of injections. Frequent treatment and monitoring schedules remain a significant burden to patients, caregivers and physicians. The proposed Phase 3 study aims to address these.


Status: Effective 

In the current study, RTH258 patients will receive q12 maintenance dosing. Disease activity assessments will be conducted by a masked investigator at Weeks 16, 20, 32 and 44, allowing four time points up to the primary endpoint of the study (Week 48) where RTH258 q12 subjects can be reassigned to q8 treatment. It is expected that early determination at Week 16 and Week 20 of subjects who are more suited to a q8 dosing regimen will minimize the percentage of q12 subjects who will require reassignment at later time points. Analyses from the PIER (Regillo 2008) and EXCITE (Schmidt-Erfurth 2011) studies have shown that visual and anatomic response during and for the 12 weeks after the loading phase are associated with visual acuity outcomes over the remainder of the first year of treatment. In addition, recent analyses from the EXCITE (Chong 2013) study have also shown that subjects who lose vision during the initial loading phase will have better visual outcomes with more frequent treatment versus q12 treatment. Finally, analyses from CATT (Kim 2014, Ying 2014) and EXCITE (Simader 2014) have also shown that new intraretinal fluid (IRF)/intraretinal cysts (IRC), and to a lesser degree CSFT increase, are associated with later visual acuity decline.

#### 5.2 Benefits and Potential Risks

RTH258 is an inhibitor of VEGF with a mechanism of action similar to ranibizumab but with a smaller molecular size (26 kDa and 48 kDa respectively).

Nonclinical studies have demonstrated that RTH258 is at least as potent as ranibizumab, with a similar vitreal half-life and a significantly lower systemic exposure. The low systemic exposure should confer a good safety profile even at a high dose. The higher dose, similar half-life, and potency of RTH258 may confer a longer treatment duration compared to currently available treatments. Two clinical studies, C-10-083 and C-12-006, have demonstrated that RTH258 is as effective as ranibizumab and aflibercept in improving BCVA outcomes whilst having a reduced treatment frequency, thus providing a potential benefit to patients and their caregivers/physicians. The ocular and systemic safety profile of single or repeated doses of RTH258 were also evaluated in the C-10-083 and C-12-006 studies, respectively, and demonstrated similar safety profiles to ranibizumab and aflibercept. Further details of the known and potential risks and benefits associated with RTH258 are presented in the Investigator's Brochure.

Summarized, the results from the Phase 2 studies demonstrate that RTH258 has similar efficacy to currently available treatment options with potentially greater duration. These data support the further development of RTH258 with a treatment regimen including q12 maintenance dosing.


Status: Effective 

#### 6 ETHICS

This clinical study will be conducted in accordance with the principles of the Declaration of Helsinki, and in compliance with the International Conference on Harmonization (ICH) E6 Good Clinical Practice (GCP) Consolidated Guideline and other regulations as applicable. The Investigator and all clinical study staff will conduct the clinical study in compliance with the protocol. The Investigator will ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience.

Before clinical study initiation, this protocol, the informed consent form (ICF), any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB). The Investigator must provide documentation of the IEC/IRB approval to the Sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), ICF, all applicable recruiting materials, written information for subject, and subject compensation programs. The IEC/IRB must be provided with a copy of the Investigator's Brochure, any periodic safety updates, and all other information as required by local regulation and/or the IEC/IRB. At the end of the study, the Investigator will notify the IEC/IRB about the study's completion. The IEC/IRB will also be notified if the study is terminated prematurely. Finally, the Investigator will report to the IEC/IRB on the progress of the study at intervals stipulated by the IEC/IRB.

Voluntary informed consent will be obtained from every subject (and/or legal representative, as applicable) prior to the initiation of any screening or other study related procedures. The Investigator must have a defined process for obtaining consent. Specifically, the Investigator, or designee, will explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved ICF. The subject must be provided an opportunity to ask questions of the Investigator, and if required by local regulation, other qualified personnel. The Investigator must provide the subject with a copy of the ICF written in a language the subject understands. The ICF must meet all applicable local laws and will provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the investigational product, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and will be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also will be told that their records may be accessed by appropriate


Status: Effective 

authorities and Sponsor designated personnel. The Investigator must keep the original, signed copy of the ICF and must provide a duplicate copy to each subject.

#### 7 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments will be created by the Sponsor and must be approved by the IEC/IRB prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the ICF and other study-related material be revised. If the ICF is revised, all subjects currently enrolled in the study may be required by the IEC/IRB to sign the approved, revised ICF.

## 8 SUBJECT POPULATION

The study population includes approximately 990 subjects to be randomized at approximately 320 sites. To participate in the study, subjects must be  $\geq$  50 years of age with untreated active CNV secondary to AMD in the study eye. The expected duration of subject participation in the randomized portion of the study is 96 weeks. The complete inclusion and exclusion criteria are presented in Section 1.

#### 9 TREATMENTS ADMINISTERED

At Visit 1/Baseline (Day 0), all eligible subjects will be randomized centrally using Interactive Response Technology (IRT) in a 1:1:1 ratio to receive either RTH258 3 mg/50  $\mu$ L, RTH258 6 mg/50  $\mu$ L, or aflibercept 2 mg/50  $\mu$ L. Randomization for subjects in Japan will be stratified according to presence or not of polypoidal choroidal vasculopathy (PCV) identified using indocyanine green (ICG) imaging and confirmed by the Central Reading Center (CRC) at the screening visit.

In the event that IRT is not available for randomization, the site should contact the Sponsor about how to proceed. In these cases subjects may be manually randomized.

Throughout the study, the Investigator will be responsible for the accounting of all study materials and investigational products, and will ensure that the investigational products are not used in any unauthorized manner.

# 9.1 Identity of Study Treatments

Test Article: RTH258 solution for IVT injection, 3 mg in 50 μL and 6 mg in 50 μL


Status: Effective 

Control Article: Aflibercept solution for IVT injection, 2 mg in 50 µL

The RTH258 trial kits will consist of a carton that contains 1 single use, sterile glass vial containing RTH258.

The availability of the control article, as well as regional regulatory requirements, will determine aflibercept sourcing. Some sites will be supplied with aflibercept by the Sponsor and others may be requested to utilize vials from their own stock.

<u>Sponsor supplied</u>: The aflibercept trial kits consist of a masked, numbered carton containing one commercially labeled vial of aflibercept.

<u>Site supplied</u>: Aflibercept will be obtained by the site in its original package. In these cases masked, numbered, empty kits will be supplied that contain instructions to administer an aflibercept injection. The lot number and expiry date of the aflibercept will be recorded.

Kit labels on all trial kits will include the kit number, protocol number, storage conditions, and a statement that the product is for investigational use only.

*All trial kits* should be stored at 2° to 8°C (35.6° to 46.4°F); do not freeze. To ensure proper conditions are maintained, a daily (7 days/week) temperature log will be maintained documenting appropriate investigational product storage conditions.

# 9.2 Usage

RTH258 3 mg and RTH258 6 mg will be administered by IVT injection. All doses will be delivered in 50  $\mu$ L (0.05 mL). Both treatment groups will receive 3 loading doses of their respective treatment at Visit 1/Day 0, Visit 2/Week 4 and Visit 3/Week 8. After the loading doses subjects will receive q12 treatment unless there is disease activity according to the guidance provided in Section 10.1. If disease activity is identified, the subject will be reassigned to receive injections q8 thereafter up to Visit 25/Week 92.

Aflibercept will be administered as a 2 mg dose in a 50  $\mu$ L (0.05 mL) injection. Subjects randomized to receive aflibercept will receive 3 loading doses at Visit 1/Day 0, Visit 2/Week 4 and Visit 3/Week 8 followed by injections at q8 intervals up to Visit 25/Week 92.

To maintain masking, beginning at Visit 6/Week 16, if a subject does not receive an active injection, they will receive a sham injection.


Status: Effective 

If at any visit, including Baseline, a subject is accidentally treated with investigational product (IP) from an arm other than the one to which they were assigned, they will be treated with the IP to which they were randomized to and according to the treatment schedule of that arm for the remainder of the study. Any instance of this must be reported to the Sponsor immediately.

## 9.3 Accountability Procedures

Each site must have designated unmasked site personnel who, upon receipt of the IP, will conduct an inventory. At the appropriate study visits, designated unmasked study staff will provide the IP to the unmasked injecting physician in accordance with the IRT procedures.

During the study, the Investigator must maintain records of IP dispensation and collection for each subject. This record must be made available to the unmasked study monitor for the purposes of verifying the accounting of clinical supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. At the conclusion of the study, the Investigator will be responsible for returning all used and unused study supplies unless otherwise instructed by the Sponsor.

## 9.4 Subject Confidentiality and Methods Used to Minimize Bias

The Investigator must ensure that the subject's anonymity is maintained throughout the course of the study. In particular, the Investigator must keep an enrollment log with confidential identifying information that corresponds to the subject number of each study participant. At the end of the clinical study, the Sponsor will collect a copy of the enrollment log without any identifying subject information. All documents submitted to the Sponsor will identify the subject exclusively by number and demographic information. No other personally identifying information should be transmitted to the Sponsor.

The intent of masking is to limit the occurrence of conscious and unconscious bias in the conduct and interpretation of the clinical study. Bias could arise from the influence that the knowledge of a specific treatment assignment may have on the recruitment and allocation of subjects, their subsequent care, the assessment of end points, the handling of withdrawals, and so on. The essential aim of masking, therefore, is to prevent identification of the treatments by the Investigator, subject, and others associated with the conduct of the study until all such opportunities for bias have passed.

This study will be double-masked, with subjects randomized to be treated with RTH258 3 mg, RTH258 6 mg or aflibercept 2 mg. All members of the Clinical Study Team will be masked to treatment assignments while the study is in progress. In addition, the biostatistician


Status: Effective 

who is directly involved in the conduct of the study (i.e. involved in patient level discussions or direct interaction with sites) will remain masked to treatment assignments while the study is in progress. Sponsor personnel who have access to treatment codes (eg, SAS® Programming, personnel directly involved with bioanalysis of serum samples, unmasked monitors performing IP accountability, and Clinical Supplies personnel) will not divulge the codes to subjects, Investigators, site staff, Sponsor Clinical Trial Management (CTM), or Sponsor Clinical Site Management (CSM). If necessary, the Sponsor may be required to unmask a subject if an adverse event (AE) meets criteria of a Suspected Unexpected Serious Adverse Reaction (SUSAR) in order to fulfill expedited regulatory reporting requirements. In this event, the Sponsor Safety Review Team will not divulge the treatment code to any other personnel involved in reporting, obtaining, and/or reviewing the clinical evaluations. This level of masking will be maintained throughout the conduct of the study.

Each site must have both masked and unmasked physicians available. The physician who performs the injection will be unmasked to the treatments as will any other site personnel who have been delegated responsibility for working with the IP. The unmasked site personnel and unmasked injecting physician must not perform BCVA, complete ophthalmic examination, disease activity assessments or administer the VFQ-25. Also, the unmasked site personnel and unmasked injecting physician must not perform assessment of any ocular or nonocular safety parameters, or assess causality AEs for subjects during the course of the study except an event reported immediately following IVT injection. The unmasked physician/site personnel should, however, assess subject safety immediately following injection (ie, they will perform the postinjection assessment; the masked physician/site personnel should not perform this assessment). Unmasked monitors will be provided to perform IP accountability.

Treatment will be assigned to subjects through the IRT system. Each subject number will be associated with treatment groups according to a random process. Subjects will be assigned treatment in numerical order; the randomization schedule will be blocked to ensure a balance of treatment allocations across the study. The IRT system will be utilized to implement the outcome of the disease activity assessments at the appropriate visits.

The randomization scheme will be generated and maintained by the Sponsor. Once all study data have been verified, validated, and the database locked, individual subjects will be unmasked to their treatment. In the event of a medical emergency during the study where the knowledge of subject treatment is required, an individual Principal Investigator will have the ability to unmask the treatment assignment for a specific subject. The Investigator should notify the Sponsor prior to unmasking a subject, if there is sufficient time. Further, the


Status: Effective 

Sponsor must be informed whenever the randomization code is broken and the reasons for unmasking.

## 10 STUDY PROCEDURES

### 10.1 Outline of Study

This is a prospective, randomized, double masked, multicenter, 3 arm study. Subjects with untreated active CNV secondary to AMD who meet all inclusion/exclusion criteria will be included in the study. The study will be conducted at approximately 320 sites and will randomize approximately 990 subjects.

The Investigator or a designee is responsible for scheduling study visits and ensuring subject compliance with the visit schedule. Subjects missing a scheduled visit should be contacted immediately to reschedule the examination, preferably within the specified study visit period.

SD-OCT imaging, fluorescein angiography (FA) and color fundus photography will be performed at the Screening Visit and the images will be assessed by CRC. In Japan, ICG will also be performed and the images will be assessed by the CRC. The CRC will review these images to confirm subject eligibility based upon the lesion attributes specified in the inclusion/exclusion criteria. Subjects who meet all inclusion and no exclusion criteria, and are confirmed as eligible by the CRC will return to the site for the Visit 1/Baseline (Day 0).

At the Visit 1/Baseline, subjects will be randomized to 1 of 3 arms in a 1:1:1 ratio per the randomization schedule.

#### **Arms 1 and 2 (RTH258):**

Subjects randomized to RTH258 3 mg (Arm 1) and RTH258 6 mg (Arm 2) will be initially injected at 4 week intervals, at Visit 1/Day 0, Visit 2/Week 4 and Visit 3/Week 8.

Following these loading doses, each subject will be injected q12 up to Week 92 unless there is disease activity according to the guidance provided at Visit 6/Week 16, Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 or Visit 22/Week 80. If disease activity is identified, the subject will be reassigned to receive injections q8 thereafter, up to Week 92. The IRT system will make the necessary changes to the dosing per the masked Investigator's assessment. The disease activity assessment will also be performed at Visit 25/Week 92 but will not be entered into IRT and will have no effect on the subject's treatment regimen.


Status: Effective 

#### Disease Activity Criteria at Week 16:

• Decrease in BCVA of  $\geq 5$  letters compared with Baseline

- Decrease in BCVA of ≥ 3 letters and CSFT increase ≥ 75µm compared with Week 12
- Decrease in BCVA of ≥ 5 letters due to neovascular AMD disease activity compared with Week 12
- New or worse IRC/IRF compared with Week 12

#### Disease Activity Criterion at Weeks 20, 32 and 44:

 Decrease in BCVA of ≥ 5 letters due to neovascular AMD disease activity compared with Week 12

#### Disease Activity Criterion at Weeks 56, 68, 80 and 92:

 Decrease in BCVA of ≥ 5 letters due to neovascular AMD disease activity compared with Week 48

A subject randomized to RTH258 who misses Visit 6/Week 16 will undergo disease activity assessment at Visit 7/Week 20 as he/she would have done if the visit had not been missed. If, however, a subject randomized to RTH258 misses any of the following disease activity assessment visits (Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 or Visit 22/Week 80) then the subject will be assumed to have met the disease activity criterion at the missed visit and will be reassigned to a q8 regimen up to study exit. The IRT system will make the necessary changes once the missed visit is registered.

If a subject misses Visit 5/Week 12, then the Visit 3/Week 8 values will be applied as the reference for disease activity assessments up to and including Visit 13/Week 44. If a subject misses Visit 14/Week 48, then the Visit 13/Week 44 values will be applied as the reference for disease activity assessments in the second year of the study.

#### Arm 3 (aflibercept 2 mg):

Subjects randomized to receive aflibercept will receive loading doses at Visit 1/Day 0, Visit 2/Week 4 and Visit 3/Week 8 followed by injections q8 thereafter up to Week 92.

Print Date:


Status: Effective 





#### 10.2 Visits and Examinations

Details of all procedures, definitions and grading criteria for test parameters can be found in the Manual of Procedures (MOP) for this protocol.

## 10.2.1 Screening Visit (Day -14 to Day -2)

The completion of assessments for this visit may occur on different days. The screening period starts with the first screening procedure (other than signing of the ICF).

One time rescreening of subjects will be allowed in the following circumstances: a) laboratory test(s) need to be repeated, b) when a subject has a temporary medical condition precluding participation. As long as testing can be repeated within 14 days of the first screening, the other screening assessments do not need to be repeated. If rescreening is to occur beyond 14 days from the original screening visit date, then all screening procedures must be repeated. Rescreening will not be permitted for the purpose of capturing new BCVA or imaging assessments that previously failed to qualify the subject. Medical judgment should be exercised to ensure that treatment is not withheld in order for a subject to participate in the study.

Explain the purpose and nature of the study, and have the subject read, sign, and date
the IRB/IEC-approved ICF. Additionally, have the individual obtaining the ICF, the
subject and a witness, if applicable, sign and date the ICF. Provide a photocopy of the
signed document to the subject and maintain the original signed document at the site.

The ICF must be signed/dated prior to performing study procedures including


Status: Effective 

#### screening.

- 2. Obtain demographic information and medical history, including information on all medications used within the past 90 days.
- 3. Perform a general physical exam.
- 4. Collect vital signs (blood pressure and pulse).
- 5. Perform a pregnancy test if the subject is female and of childbearing potential.
- 6. Obtain blood and urine samples for blood chemistry/hematology and urinalysis and forward the samples to the central laboratory. *Blood draws should be performed prior to injection of fluorescein dye*.
- 7. Perform BCVA on both eyes.
- 8. Perform a complete ophthalmic examination on **both eyes** including slit-lamp exam, intraocular pressure (IOP) measurement and fundus exam.
- 9. Perform SD-OCT on **both eyes**. Submit the images (within 24 hours, if possible) to the CRC for determination of eligibility.
- 10. Perform FA on **both eyes**. Submit the images (within 24 hours, if possible) to the CRC for determination of eligibility.
- 11. Perform 3-field color fundus photography on **both eyes**. Submit the images (within 24 hours, if possible) to the CRC for determination of eligibility.
- 12. **At Japanese sites**: Perform ICG imaging on **both eyes**. Submit the images (within 24 hours, if possible) to the CRC for AMD subtype analysis.
- 13. Register the subject (including screen fails) in the Electronic Data Capture (EDC) system and obtain a subject ID number.
- 14. Contact IRT to enter the subject ID number.
- 15. Monitor for AEs.
- 16. Schedule Visit 1/Baseline to take place 2 to 14 days after the start of the Screening assessments.


Status: Effective 

## 10.2.2 Visit 1/Baseline (Day 0)

At the Baseline Visit, subjects will be randomized only if the subject has successfully met all of the eligibility criteria.

- 1. Obtain information on any changes in medical health and/or the use of concomitant medications.
- 2. Record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing.
- 3. Administer the VFQ-25, using validated translations as applicable and available. The VFQ-25 should be administered prior to any examination.
- 4. Collect vital signs (blood pressure and pulse).
- 5. Obtain a blood sample for anti-drug antibody (ADA) analysis. *Blood draws should* take place prior to the IVT injection.
- 6. Obtain a blood sample for systemic RTH258 analysis. *Blood draws should take place prior to the IVT injection.*
- 7. Perform BCVA on **both eyes.** Baseline BCVA of the study eye must be between 78 and 23 letters, inclusive, for the subject to qualify.
- 8. Perform a complete ophthalmic examination on the **study eye** including slit-lamp exam, IOP measurement, and fundus exam (dilation to be performed at the discretion of the Investigator).
- 9. Perform SD-OCT imaging on the **study eye** and submit the images to the CRC.
- 10. Where applicable, perform fundus autofluorescence (FAF) imaging on the **study eye** and submit the images to the CRC. *FAF will only be performed at a subset of sites*.
- 11. Verify that all eligibility criteria have been met, including the required screening imaging eligibility from the CRC. The Investigator should also review the results from the central laboratory for the samples collected at Screening to determine if there is anything that would preclude participation of the subject.
- 12. Contact IRT to obtain a kit number.
- 13. Have the unmasked Investigator perform an IVT injection according to the


Status: Effective 

randomization/kit assignment. The injection procedure may be performed at a later time, as long as it occurs within 7 days of the scheduled visit.

- 14. After the injection, perform a postinjection assessment of the **study eye** 0-5 minutes and at 30 ( $\pm$  15) minutes after injection (and at further time points, as needed).
- 15. Schedule Visit 2/Week 4 to take place  $28 \pm 3$  days after Visit 1/Baseline.

# 10.2.3 Visit 2/Week 4 (Day 28 ± 3 Days) and Visit 3/Week 8 (Day 56 ± 3 Days)

- 1. Obtain information on any changes in medical health and/or the use of concomitant medications.
- 2. Record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing.
- 3. Collect vital signs (blood pressure and pulse).
- 4. Obtain a blood sample for ADA analysis (*Visit 2 only*). Blood draws should take place prior to the IVT injection.
- 5. Obtain a blood sample for systemic RTH258 analysis (*Visit 2 only*). *Blood draws should take place prior to the IVT injection*.
- 6. Perform BCVA on the **study eye.**
- 7. Perform a complete ophthalmic examination on the **study eye** including slit-lamp exam, IOP measurement, and fundus exam (dilation to be performed at the discretion of the Investigator).
- 8. Perform SD-OCT imaging on the **study eye** and submit the images to the CRC.
- 9. Contact IRT to obtain a kit number.
- 10. Have the unmasked Investigator perform an IVT injection according to the randomization/kit assignment. The injection procedure may be performed at a later time, as long as it occurs within 7 days of the scheduled visit and is within the visit window.
- 11. After the injection perform a postinjection assessment of the **study eye** 0-5 minutes


Status: Effective 

and at 30 ( $\pm$  15) minutes after injection (and at further time points, as needed).

12. Schedule Visit 5/Week 12 to take place  $84 \pm 7$  days after Visit 1/Baseline.

## 10.2.4 Visit 4 (Visit 3 + 1 Day)

This visit only applies to the subset of subjects who were randomly selected to attend it and did so before Version 3.0 of the protocol became effective.

# 10.2.5 Visit 5 /Week 12 (Day $84 \pm 7$ Days) Through Visit 25 /Week 92 (Day $644 \pm 7$ Days)

- 1. Obtain information on any changes in medical health and/or the use of concomitant medications.
- 2. Record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing.
- 3. Administer the VFQ-25, using validated translations as applicable and available (*Visit 8, Visit 14 and Visit 20 only*). The VFQ-25 should be administered prior to any examination.
- 4. Perform a general physical exam. (Visit 14 only).
- 5. Collect vital signs (blood pressure and pulse).
- 6. Perform a pregnancy test if the subject is female and of childbearing potential (*Visit 14 only*).
- 7. Obtain blood and urine samples for blood chemistry/hematology and urinalysis and forward the samples to the central laboratory (*Visit 5 and Visit 14 only*). Blood draws should be performed prior to any IVT or sham injection and prior to injection of fluorescein dye.
- 8. Obtain a blood sample for ADA analysis (*Visit 5, Visit 8, Visit 11, Visit 14, Visit 19, Visit 24 only*). Blood draws should be performed prior to any IVT or sham injection and prior to any injection of fluorescein dye.


Status: Effective 

9. Obtain a blood sample for systemic RTH258 analysis (*Visit 5, Visit 8, Visit 11, Visit 14, Visit 19, Visit 24 only*). Blood draws should be performed prior to any IVT or sham injection and prior to any injection of fluorescein dye.

10. Perform BCVA on the study eye.

Perform BCVA on both eyes (Visit 5, Visit 8, Visit 11, Visit 14, Visit 17, Visit 20 and Visit 23 only).

11. Perform a complete ophthalmic examination on the **study eye** including slit-lamp exam, IOP measurement and fundus exam (dilation to be performed at the discretion of the Investigator).

Perform a complete ophthalmic exam on both eyes (Visit 14 only).

- 12. Perform SD-OCT on the **study eye** and submit the images to the CRC.

  Perform SD-OCT on **both eyes** and submit the images to the CRC (*Visit 14 only*).
- 13. Perform FA (**study eye** only at Visit 5, **both eyes** at Visit 14) and submit the images to the CRC (*Visit 5 and Visit 14 only*).
- 14. Perform color fundus photography (**study eye** only at Visit 5, **both eyes** at Visit 14) and submit the images to the CRC (*Visit 5 and Visit 14 only*).
- 15. Where applicable, perform FAF imaging on the **study eye** and submit the images to the CRC (*Visit 5 and Visit 14 only*). FAF will only be performed at a subset of sites.
- 16. Have the masked Investigator perform the visit appropriate disease activity assessment for the study eye (Visit 6, Visit 7, Visit 10, Visit 13, Visit 16, Visit 19, Visit 22 and Visit 25 only).
- 17. Contact IRT (all visits except Visit 5).
- 18. Have the unmasked Investigator perform an IVT or sham injection according to the randomization/kit assignment (all visits except Visit 5). The injection procedure may be performed at a later time, as long as it occurs within 7 days of the scheduled visit and is within the visit window.
- 19. After injection perform a postinjection assessment of the **study eye** 0-5 minutes and at 30 ( $\pm$  15) minutes (and at further time points, as needed) (all visits except Visit 5).
- 20. Schedule Visit 26/Week 96 to take place  $672 \pm 7$  days after Visit 1/Baseline.


Status: Effective 

## 10.2.6 Visit 26/Week 96/Exit Visit (Day $672 \pm 7$ Days) or Early Exit

- 1. Obtain information on any changes in medical health and/or the use of concomitant medications.
- 2. Record any AEs that are observed or reported, including those associated with changes in concomitant medication dosing.
- 3. Administer the VFQ-25, using validated translations as applicable and available. The VFQ-25 should be administered prior to any examination.
- 4. Perform a general physical exam.
- 5. Collect vital signs (blood pressure and pulse).
- 6. Perform a pregnancy test if the subject is female and of childbearing potential.
- 7. Obtain blood and urine samples for blood chemistry/hematology and urinalysis and forward the samples to the central laboratory. *Blood draws should be performed prior to injection of fluorescein dye*.
- 8. Obtain a blood sample for ADA analysis (if the subject exits at or before Visit 24).

  Blood draws should be performed prior to injection of fluorescein dye.
- 9. Obtain a blood sample for systemic RTH258 analysis (if the subject exits at or before Visit 24). Blood draws should be performed prior to injection of fluorescein dye.
- 10. Perform BCVA on both eyes.
- 11. Perform a complete ophthalmic examination on **both eyes** including slit-lamp exam, IOP measurement and fundus exam (dilation to be performed at the discretion of the Investigator).
- 12. Perform SD-OCT imaging on **both eyes** and submit the images to the CRC.
- 13. Perform FA on **both eyes** and submit the images to the CRC.
- 14. Perform color fundus photography on **both eyes** and submit images to the CRC.
- 15. Where applicable, perform FAF on the **study eye** and submit the images to the CRC. *FAF will only be performed at a subset of sites*.
- 16. Complete the Exit Form.


Status: Effective 

#### 10.3 Unscheduled Visits

If a subject returns to the site prior to their next scheduled study visit for assessment of an adverse event, the Unscheduled Visit pages of the electronic case report form (CRF) should be completed. Procedures conducted at the Unscheduled Visit are at the discretion of the Investigator apart from treatments of the study eye for AMD. If the subject is discontinuing at the Unscheduled Visit, the CRFs for the Exit Visit should be completed rather than the CRFs for an Unscheduled Visit. Routine treatments and routine follow-up of the nonstudy eye will not be considered an Unscheduled Visit. Any treatments of the nonstudy eye will be captured on the Concomitant Medication Page.

## 10.4 Discontinued Subjects

Discontinued subjects are those who are lost to follow-up, withdraw or are withdrawn from the study after the Visit 1/Baseline. Subjects may discontinue from the study at any time for any reason. Discontinued subjects will not be replaced (ie, their subject numbers will not be re-assigned/re-used). The site must contact IRT to register the subject's discontinuation from IP.

Should a subject exhibit any clinically relevant signs, symptoms, or other clinical observations that possibly could be associated with suspected sensitivity or intolerance to one of the study treatments, the Investigator must document those observations on an AE Form (AEF). If a subject discontinues the study with an ongoing AE, follow-up procedures, as appropriate and outlined in Section 12.6, should be performed.

Any subject who exits early from the study must undergo all procedures outlined at Visit 26/Week 96 (Section 10.2.6). Additionally, the Exit Form must be completed and a reason for discontinuation must be identified.

If a subject exits early from the study between visits, the Investigator must attempt to contact the subject and request the subject to return for a final visit to complete the exit procedures. If the subject is unable or unwilling to return for the Exit Visit, the subject will be considered lost to follow-up and the 'date of exit' will be the date that the subject was last seen at the site or contacted by other communication.

Finally, to ensure the safety of all subjects who exit early from the study, Investigators should assess each subject and, if necessary, advise them of any therapies and/or medical procedures that might be needed to maintain their health.


Status: Effective 

## 10.5 Discontinuation of Study Treatment

The Investigator may discontinue study treatment for a given subject and/or withdraw the subject from study if he/she believes that continuation would pose a risk to their health.

Subjects can be discontinued from study treatment because of:

- appearance of a new health condition suspected to require appropriate care or require medications prohibited by the protocol
- refusal to continue treatment, or at the Investigator's discretion based on his/her clinical judgment the subject requires rescue treatment
- use of prohibited treatment during the study
- investigator's discretion based on his/her clinical judgment
- positive urine/serum pregnancy test

Subjects who discontinue study treatment should NOT be considered withdrawn from the study. Subjects are expected to continue with the study visits and procedures as long as such procedures do not pose a risk to the well-being of the subject. Site personnel must also contact IRT to register the subject's discontinuation from study treatment.

The appropriate personnel from the site and Sponsor will assess whether study treatment should be discontinued for any subject whose treatment code has been broken inadvertently for any reason.

## 10.6 Clinical Study Termination

If the clinical study is prematurely terminated or suspended, the Sponsor will inform the Investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension. The Investigator should promptly notify the IEC/IRB of the termination or suspension and of the reason(s). The Sponsor reserves the right to close the investigational site or terminate the study in its entirety at any time, for reasonable cause. Reasons for the closure of an investigational site or termination of a study may include:

- The Investigator fails to comply with the protocol or GCP guidelines
- Safety concerns
- Sufficient data suggesting lack of efficacy


Status: Effective 

Inadequate recruitment of subjects by the Investigator

The Investigator also may terminate the study at his/her site for reasonable cause. If the Sponsor terminates the study for safety reasons, it will immediately notify the Investigator(s) by telephone and subsequently will provide written confirmation of and instructions for study termination. The investigator may be informed of additional procedures to be followed in order to ensure that adequate consideration is given to the protection of the patient's interests. The investigator will be responsible for informing the IRBs/IECs of the early termination of the trial.

### 10.7 Study Methods and Measurements

## 10.7.1 Visual Function Questionnaire-25

Quality of life data will be collected with a visual function questionnaire using the National Eye Institute VFQ-25 which is a validated instrument that has been used in many studies of subjects with AMD. The VFQ-25 will be administered by masked site staff to subjects at sites where local language versions are available, validated, and approved by the IEC/IRB. The VFQ-25 must be administered before any other examination. The United States English version of the VFQ-25 is included in the MOP.

## 10.7.2 General Physical Exam and Vital Signs

The physical exam will consist of a routine evaluation of organ systems eg., ears, eyes, nose, throat, neck, lymph nodes, lungs, heart, abdomen, skin/extremities, neurological, and musculoskeletal systems. After Screening, the physical exam will also include a discussion with the subject if there have been changes in his/her physical condition since the Screening exam. All clinically significant findings will be recorded as medical history or adverse events, as appropriate.

Vital signs consist of blood pressure and pulse rate measurements. Standardized procedures for each are provided in the MOP.

# 10.7.3 Pregnancy Test

A pregnancy test will be conducted for all women of child bearing potential at Screening, Visit 14/Week 48, and Exit Visit. Urine pregnancy tests will be performed unless local regulations require serum pregnancy tests. Additional pregnancy testing may be conducted at the Investigator's discretion or if required by local regulations.


Status: Effective 

### 10.7.4 Laboratory Analysis of Blood and Urine

Blood and urine samples will be shipped to a central laboratory. Results of the analysis will be provided to the Investigator who will assess those from Screening prior to randomizing the subject to determine if there is anything that would preclude participation of the subject and at subsequent visits to assess any changes from Screening. A standardized procedure for the collection and processing of blood and urine is provided in a separate laboratory hand book. A list of laboratory parameters is provided in the MOP. If a subject should present with a clinically significant change resulting in an adverse event, as assessed by the Investigator, a decision will be made as to subject continuation in the trial. This decision will take into account the adverse event characteristics including but not limited to seriousness and relationship to study drug.

# 10.7.5 Analysis of Anti-drug Antibodies (ADA) and Systemic RTH258

Collection of blood for ADA and systemic RTH258 should take place prior to any injection/sham. A standardized procedure for the collection, processing, storage and shipment of these blood samples is provided in a separate laboratory hand book.

## 10.7.6 Best-Corrected Visual Acuity

ETDRS visual acuity testing should precede any examination requiring administration of eye drops to dilate the eye or any examination requiring contact with the eye. Visual acuity testing should be performed following refraction and completed according to the procedure outlined in the MOP. Certification of the facility, equipment and examiners at each investigative site will occur prior to any evaluation of study subjects.

Subjects at sites in Japan and some Asian countries will undergo BCVA testing using numerical charts rather than letter charts. Therefore, all references in the protocol to changes in letters read will be changes in numbers in these countries.

# 10.7.7 Complete Ophthalmic Examination

A complete description of standardized procedures and grading scales is outlined in the MOP. The ophthalmic exam will consist of the following:

 Slit-lamp examination – includes evaluation of the lids/lashes, conjunctiva, cornea, iris, lens, and aqueous reaction (cells and flare).


Status: Effective 

 IOP measurement – a measurement of intraocular pressure will be conducted using an applanation tonometer or Tonopen. The same method should be used throughout the study for each subject.

 Fundus exam – includes evaluation of the vitreous, retina, macula, choroid, and optic nerve. Dilation for the fundus exam is at the discretion of the Investigator.

## 10.7.8 Spectral Domain Optical Coherence Tomography Imaging

A standardized procedure for the collection of quantitative and qualitative data via SD-OCT is provided by the CRC in a separate hand book. Each site must select a single brand of equipment for use on all subjects at that site. Certification of the equipment and examiners at each investigative site will occur prior to evaluation of study subjects. At the Screening Visit, SD-OCT images will be submitted to the CRC for determination of eligibility. Feedback from the CRC following expedited review will be provided to the sites via email or fax. The CRC may participate in the assessment of new disease activity, as appropriate.

### 10.7.9 Fluorescein Angiography

A standardized procedure for the collection of FA images is provided by the CRC in a separate hand book. Certification of the equipment and examiners at each investigative site will occur prior to evaluation of study subjects. At the Screening Visit, retinal images will be submitted to the CRC for determination of eligibility. FA images from previous routine evaluations may be used as long as they were performed within 3 days of the Screening Visit using CRC-certified equipment and examiners. Feedback from the CRC following expedited review will be provided to the sites via email or fax.

# 10.7.10 Color Fundus Photography

A standardized procedure for the collection of 3-field color fundus photographic images is provided by the CRC in a separate hand book. Certification of the equipment and examiners at each investigative site will occur prior to evaluation of study subjects. At the Screening Visit retinal images will be sent to the CRC for determination of eligibility. Feedback from the CRC following expedited review will be provided to the sites via email or fax.

# 10.7.11 Indocyanine Green

At all sites in Japan, ICG images will be taken at Screening. A standardized procedure for the collection of ICG images is provided by the CRC in a separate hand book. Certification of the equipment and examiners at each investigative site will occur prior to evaluation of study subjects. At the Screening Visit, ICG images will be sent to the CRC for determination of


Status: Effective 

AMD subtype which will be provided following expedited review and will be utilized by IRT in the randomization process.

#### **10.7.12** Fundus Autofluorescence

FAF will be performed at a subset of sites in order to assess the occurrence of geographic atrophy. A standardized procedure for the collection of FAF images is provided by the CRC in a separate hand book. Certification of the equipment and examiners at each investigative site will occur prior to evaluation of study subjects. FAF will not be used to determine eligibility, but will be included beginning at the Visit 1/Baseline.

### 10.7.13 Disease Activity Assessment

The masked Investigator will assess the study eye of all subjects at Visit 6/Week 16, Visit 7/Week 20, Visit 10/Week 32, Visit 13/Week 44, Visit 16/Week 56, Visit 19/Week 68 and Visit 22/Week 80. The IRT system will make the necessary changes to the dosing per the masked Investigator's assessment. The disease activity assessment will also be performed at Visit 25/Week 92, but will not be entered into IRT and will have no effect on the subject's treatment regimen. Details of the disease activity assessments are further outlined in the MOP.

## 10.7.14 Intravitreal Administration of Investigational Product

The IVT injection procedure for both the test article and control article is the same as that described for aflibercept in the product information sheet. IVT injection is contraindicated in subjects with active ocular or periocular infections and in subjects with active intraocular inflammation; therefore, the Investigator should verify that these conditions are not present in either eye (study and nonstudy eyes) prior to every injection. Specific instructions for injection procedures are provided in the MOP.

# 10.7.15 Administration of Sham Injection

Beginning at Visit 6/Week 16, at visits when subjects do not receive an active injection, they will be administered a sham injection. For the sham injection the tip of an injection syringe (the hub without a needle) will be used. A standardized procedure for the sham is described in the MOP.

# 10.7.16 Postinjection Assessment

The study eye will be assessed before, immediately (0-5 minutes) after and 30 ( $\pm$  15) minutes after each IVT/sham injection to ensure that the procedure and/or the study medication have


Status: Effective 

not endangered the health of the eye. The postinjection assessments include an evaluation of central retinal artery perfusion via a gross assessment of vision (e.g. count fingers) and measurement of IOP according to the schedule detailed in the MOP. Direct visualization to assess the central retinal artery, presence of retinal detachment, presence of new intraocular hemorrhage(s) might be appropriate at the discretion of the investigator and/or based on the results of gross assessment of vision and IOP measurement. Assessments will continue until the central retinal artery is adequately perfused and the IOP is within 10 mmHg of the pre-injection value and is stable in the opinion of the Investigator. Any subject who develops significantly raised IOP (> 30 mmHg) or a non-adequately perfused central retinal artery at any time during the study should be monitored according to the Investigator's clinical judgment and may undergo additional procedures and measurements of IOP beyond those specified in the protocol. If, at the conclusion of the required evaluation period following an injection/sham, there are no safety concerns, the subject will leave the site. If any concern or immediate toxicity is noted, the subject will remain at the site and will be treated according to the designated evaluating physician's clinical judgment. If any issues regarding IOP were noted during the postinjection assessment, then the subject should be scheduled for a follow-up visit (Unscheduled Visit) the day following injection/sham, if required in the opinion of the Investigator. Clinically relevant changes that are observed during the postinjection assessment should be reported as adverse events.

#### 10.8 Concomitant Treatment

The Investigator should instruct the subject to notify the study site about any new medications he/she takes after enrolling into the study.

Should the nonstudy eye require treatment during the study with an anti-VEGF, a drug which is approved for the treatment of exudative AMD in the respective country should be applied at the discretion of the Investigator and following the procedures established at the respective site. The nonstudy eye treatment may occur at any time once the Baseline study eye injection has been administered.

#### 10.9 Prohibited Treatment

Use of treatments, as displayed in Table 10-1, are not allowed after the start of the study i.e., Screening. In addition, there are certain washout periods to be respected as outlined in the exclusion criteria.


Status: Effective 

#### Table 10-1 Prohibited Medication

Medication

Study eye: Intra- or periocular corticosteroids

Study eye: Laser treatment for AMD

Study eye: Anti-VEGF therapy other than IP

Nonstudy eye: Unapproved or investigational treatment

Systemic: Systemic corticosteroids for 30 or more consecutive days (low stable doses of corticosteroids [defined as  $\leq$ 10 mg prednisolone or equivalent dose], inhaled, nasal or dermal steroids are permitted)

Systemic: Anti-VEGF therapy

Any investigational drug, biologic or device (with the exception of over-the-counter vitamins, supplements or diets)

#### 11 ANALYSIS PLAN

#### 11.1 General Considerations

Continuous variables will be summarized for the measured values and change from Baseline values using the number of observations, mean, standard deviation, median, quartiles, minimum and maximum. Categorical variables will be summarized with numbers and percent from each category. Treatment differences will be presented together with 95% confidence intervals as appropriate.

# 11.2 Subject Evaluability

Subject evaluability based on pre-specified deviations and their impact on analysis sets will be determined prior to breaking the masked treatment assignment code and locking the database for the primary analysis at Week 48. Protocol deviations and their impact on analysis sets will be pre-specified in the deviations and evaluability plan (DEP).

# 11.3 Analysis Sets

The following analysis sets are defined:

**All-enrolled analysis set**: includes all subjects who signed an ICF and are assigned subject numbers. This analysis set will be used to summarize subject disposition and pre-treatment adverse events.


Status: Effective 

**All-randomized analysis set**: includes all subjects who were randomized. This analysis set will be used to describe the randomized study population based on demographics and baseline characteristics.

**Safety analysis set**: includes all subjects who received at least one IVT injection. Subjects in the safety analysis set will be analyzed according to the first treatment received. This analysis set will be used for all safety analyses.

**Full analysis set (FAS):** includes all subjects who are randomized and received at least one IVT injection. Following the intent-to-treat (ITT) principle, subjects in the FAS will be analyzed according to the treatment group they are assigned at randomization. The FAS will be the primary analysis set for efficacy analyses.

The per protocol analysis set (PPS): defined for the primary and key secondary efficacy analysis at Week 48 includes all subjects in the FAS with no protocol deviations that are expected to majorly affect the assessment of efficacy at Week 48 including: lack of compliance (including treatment misallocation), missing data, concomitant medication and deviation from inclusion/exclusion criteria. Discontinuation from treatment due to lack of efficacy does not constitute a reason for exclusion from the PPS.Before the Week 48 database lock the relevant protocol deviations will be specified in the DEP document and identified at the subject level in the database.

## 11.4 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized for all analysis sets. All summaries will be presented by treatment group and overall.

# 11.4.1 Demographic Characteristics

The demographic parameters are age category (50 to 64, 65 to 74, 75 to 84, and  $\geq$  85), gender, ethnicity and race. Age will also be summarized as a continuous variable.

#### 11.4.2 Baseline Characteristics

Baseline characteristics will include: primary diagnosis of neovascular AMD, time since diagnosis of neovascular AMD (days), whether neovascular AMD is unilateral or bilateral, BCVA (both as a continuous variable and using categories ( $\leq 55$ , 56-70,  $\geq 71$  letters), lesion type (predominantly classic, minimally classic, pure occult), foveal involvement (subfoveal, extrafoveal, undeterminable), CNV lesion size, presence of subretinal fluid, presence of intraretinal fluid/cyst, presence of sub RPE fluid, neurosensory retinal thickness, CSFT (both as a continuous variable and using categories ( $< 400 \geq 400 \, \mu m$ ).


Status: Effective 

### 11.5 Primary and Key Secondary Efficacy Analyses

#### **Primary Efficacy Endpoint:**

Change in BCVA from Baseline to Week 48

#### **Key Secondary Efficacy Endpoints:**

- Average change in BCVA from Baseline over the period Week 36 through 48. For each subject, this endpoint is defined as the average of the changes from Baseline to Weeks 36, 40, 44 and 48
- q12 treatment status at Week 48 (for subjects randomized to RTH258 3 mg and 6 mg only)
- q12 treatment status at Week 48 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg only).

The primary and key secondary endpoints will be analyzed based on the FAS with last-observation-carried-forward (LOCF) imputation of missing BCVA values (primary and first key secondary endpoint) and a negative q12 treatment status at Week 48 in case of incomplete active treatment up to Week 48 (second and third key secondary endpoint).

## 11.5.1 Statistical Hypotheses

The statistical hypotheses for the primary endpoint and first key secondary endpoint are to demonstrate noninferiority of RTH258 3 mg and 6 mg to aflibercept 2 mg within a margin of 4 letters.

The following 4 hypotheses will be tested in the pre-specified hierarchical sequence according to their numbering (HAn, n=1,2,3,4). Consequently, confirmatory testing of a given hypothesis requires rejection of all preceding null hypotheses. In this setting, each hypothesis will be assessed at a two-sided significance level of 0.05, while keeping the global type I error rate at 0.05.

**Hypotheses**: The following noninferiority hypotheses are related to a noninferiority margin of 4 letters.

 $_{48}$  = Week 48,  $_{36-48}$  = Week 36 through 48,  $_{R6(3)}$ =RTH258 6(3) mg,  $_{A}$ =Aflibercept 2 mg


Status: Effective 

**H**<sub>01</sub>:  $\mu_{48R6}$  -  $\mu_{48A} \le -4$  letters vs **H**<sub>A1</sub>:  $\mu_{48R6}$  -  $\mu_{48A} > -4$  letters

**H**<sub>02</sub>:  $\mu_{36-48R6}$  -  $\mu_{36-48A} \le -4$  letters vs **H**<sub>A2</sub>:  $\mu_{36-48R6}$  -  $\mu_{36-48A} \ge -4$  letters

 $\mathbf{H}_{03}$ :  $\mu_{48R3}$  -  $\mu_{48A} \le -4$  letters vs  $\mathbf{H}_{A3}$ :  $\mu_{48R3}$  -  $\mu_{48A} > -4$  letters

 $\mathbf{H_{04}}$ :  $\mu_{36\text{-}48R3}$  -  $\mu_{36\text{-}48A} \le$  -4 letters vs  $\mathbf{H_{A4}}$ :  $\mu_{36\text{-}48R3}$  -  $\mu_{36\text{-}48A} >$  -4 letters

 $\mu_{48R6}$ ,  $\mu_{48R3}$  and  $\mu_{48A}$  being the corresponding unknown true mean BCVA changes from Baseline to Week 48.

 $\mu_{36\text{-}48R6}$ ,  $\mu_{36\text{-}48R3}$  and  $\mu_{36\text{-}48A}$  being the corresponding unknown true mean values for the average change in BCVA from Baseline over the period Week 36 through 48.

#### 11.5.2 Statistical Methods

For the test of noninferiority, a two-sided 95% confidence interval for the treatment difference will be derived from an analysis of variance (ANOVA) model with treatment, baseline BCVA categories ( $\leq 55$ , 56-70,  $\geq 71$  letters) and age categories (< 75,  $\geq 75$  years) as fixed effects. In order to demonstrate noninferiority, the lower limit of the two-sided 95% confidence interval for the treatment difference (RTH258 – aflibercept) must be greater than -4 letters representing the noninferiority margin.

The q12 treatment status at Week 48 in the RTH258 treatment arms will be presented descriptively together with exact 95% confidence intervals for the proportion of subjects with a positive status:

- For the (overall) proportion of subjects with a positive q12 treatment status at Week 48, the denominator is all FAS subjects in the RTH258 3 mg/6 mg groups, and the numerator is the corresponding number of subjects with no identified q8-need at Week 16, 20, 32 and 44 (while missing the Week 16 assessment is considered as no q8 treatment needed)
- For the predictability of the adequacy of q12 treatment based on the absence of disease activity during the first q12 cycle, the denominator is all FAS subjects in the RTH258 3 mg/6 mg groups with no identified q8-need at Week 16 and Week 20 (while missing the Week 16 assessment is considered a no-q8 treatment needed), and the numerator is the corresponding number of subjects with a positive q12 treatment status at Week 48 ie. with no identified q8-need at Week 16, 20, 32 and 44.


Status: Effective 

### 11.5.3 Sensitivity Analyses

Sensitivity analysis to explore the robustness of the primary efficacy results with respect to protocol deviations will use the PPS with LOCF imputation of missing values using the same model and factors as in the primary efficacy analysis model.

Sensitivity analyses to explore the robustness of the primary and first key secondary efficacy analysis results related to missing values will be performed on the observed data in the FAS applying the specified ANOVA model and a mixed model repeated measures (MMRM).

### 11.5.4 Subgroups

The following subgroups will be analyzed for the primary and key secondary efficacy endpoints:

- Age category (< 75 years and ≥75 years)</li>
- Gender (male and female)
- Baseline BCVA categories (≤ 55, 56-70, ≥ 71 letters)
- Baseline CSFT category ( $< 400, \ge 400$ )
- Baseline lesion type (predominantly classic, minimally classic, pure occult)
- Baseline lesion size (tertiles) by lesion type (predominantly classic vs. minimally classic/occult)

## 11.6 Additional Secondary Efficacy Analyses

The following secondary efficacy endpoints will be analyzed primarily based on FAS:

- Change in BCVA from Baseline to each postbaseline visit
- Average change in BCVA from Baseline over the period Week 84 through Week 96
- Average change in BCVA from Baseline over the period Week 4 to Week 48/96
- Average change in BCVA from Baseline over the period Week 12 to Week 48/96
- Gain in BCVA of 15/10/5 letters or more from Baseline to each postbaseline visit
- Loss in BCVA of 15/10/5 letters or more from Baseline to each postbaseline visit

Print Date: Print Date:


Status: Effective 

q12 treatment status at Week 96 (for subjects randomized to RTH258 3 mg and 6 mg only)

- q12 treatment status at Week 96 within the subjects with no q8 need during the first q12 cycle (Week 16, Week 20) (for subjects randomized to RTH258 3 mg and 6 mg only)
- Change in CSFT from Baseline to each postbaseline visit
- Change in neurosensory retinal thickness from Baseline to each postbaseline visit
- Change in CNV lesion size from Baseline to Weeks 12, 48 and 96
- Absence of subretinal fluid at each postbaseline visit
- Absence of intraretinal fluid at each postbaseline visit
- Absence of sub RPE fluid at each visit
- q8-treatment need status assessed at Weeks 16, 20, 32, 44, 56, 68, 80 and 92
- Change in patient-reported outcomes (VFQ-25) total and subscale scores from Baseline to Weeks 24, 48, 72 and 96

Statistical methods for the analysis of each of the secondary endpoints will be described in the statistical analysis plan (SAP).

## 11.7 Handling of Missing Data

The primary presentation of efficacy results will use LOCF for the imputation of missing values supplemented by presentations on the observed data only. All non-missing post-baseline values including assessments done at unscheduled visits will be used when implementing the LOCF imputation. Imputations related to the evaluation of the q12-treatment status at Week 96 will follow the concept described for Week 48.

# 11.8 Multiplicity

No alpha adjustment will be applied for testing the hypotheses for the primary and first key secondary efficacy analyses as the four hypotheses will be tested in the pre-specified hierarchical sequence according to their numbering. Consequently, confirmatory testing of a given hypothesis requires rejection of all preceding null-hypotheses. In this setting each

Print Date:


Status: Effective 

hypothesis will be assessed at a two-sided  $\alpha = 0.05$ , while keeping also the global type I error rate at 0.05. Other key secondary endpoints are not associated with hypothesis testing.

## 11.9 Safety

### 11.9.1 Treatment Exposure

The extent of treatment exposure will be presented based on the overall number of injections, the number of subjects injected per visit, and frequency of the different treatment patterns.

## 11.9.2 Medical History

Relevant medical history (ocular and nonocular) will be tabulated by system organ class and preferred term of the MedDRA dictionary. Ocular events will be presented by study and nonstudy eye.

## 11.9.3 Concomitant Therapies

The number and percentage of subjects taking concomitant therapies will be summarized by preferred term according to the WHO Drug Reference List dictionary. Ocular therapies will be presented by study and nonstudy eye.

## 11.9.4 Safety Parameters

The following safety parameters will be descriptively analyzed to assess treatment emergent changes or changes specifically related to the injection procedure using postinjection assessments:

- Adverse events
- General physical exam
- Vital signs
- Laboratory tests (blood chemistry, hematology and urinalysis)
- Worsening in BCVA
- Slit-lamp examination
- Fundus exam
- IOP

Print Date: Print Date:

Status: Effective 

Postinjection assessment

ADA levels

Systemic RTH258 levels

## 11.9.5 Adverse Events

AEs will be coded using the MedDRA dictionary and presented by system organ class and preferred term. Treatment emergent AEs will be analyzed based on the number and percentage of subjects with at least one AE in the category of interest. Separate presentations will be provided related to ocular events in the study eye and nonstudy eye and non-ocular events. Additional summaries will be provided by severity and causality (separately assessed for the injection procedure and the drug). Serious adverse events and adverse events leading to discontinuation of study treatment will also be summarized separately.

Subject listings of all adverse events will be provided. Deaths and other serious or clinically significant non-fatal adverse events will be listed separately.

Events of special interest (ESIs; as defined in section 12.3) will be presented based on their incidences.

## 11.10 Interim Analyses

The primary efficacy analysis will be based on the Week 48 data. The database including all Week 48 data will be locked once all active subjects have completed the Week 48 Visit. Systemic RTH258 and ADA data up to Week 36 will be analyzed for the Week 48 primary analysis. The primary analysis at Week 48 will be performed with an unmasking of specified individuals from the Sponsor who are not involved in the direct conduct of the trial.

Subjects will remain in the study and will continue to receive masked treatment through the planned duration (96 Weeks) to allow for further masked evaluation of efficacy and safety.

Treatment masking of individual subjects will remain intact for all subjects, Investigators, and staff from the Sponsor who have contact with subjects or Investigators or those who are involved in the direct conduct of the study until the final database lock has occurred.

# 11.11 Sample Size Justification

A sample size of 297 subjects per treatment arm is sufficient to demonstrate noninferiority (margin = 4 letters) of RTH258 3 mg/6 mg versus aflibercept 2 mg with respect to the BCVA

Print Date:


Status: Effective 

change from Baseline to Week 48 at a two-sided alpha level of 0.05 with a power of approximately 90% assuming equal efficacy and a common standard deviation of 15 letters. A power of at least 90% can be expected for the first key secondary endpoint assuming that averaging over the 4 time points will not lead to an increase in the standard deviation.

To account for a drop-out rate of 10%, a total of 330 subjects will be randomized per treatment arm.

### 12 ADVERSE EVENTS

### 12.1 General Information

An AE is any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, can be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. In clinical studies, any AE can include an untoward medical occurrence occurring at any time, including run-in or washout periods, even if no study treatment has been administered. The determination of clinical relevance is based upon the medical judgment of the Investigator.

## 12.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the Investigator should inquire about AEs by asking the standard questions:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take since your last study visit?"

AEs should be reported for any clinically relevant change in concomitant medication(s) that is the result of an untoward (unfavorable and unintended) change in a subject's medical health.

Changes in any protocol-specific parameters and questionnaires (if applicable) evaluated during the study are to be reviewed by the Investigator. Any untoward (unfavorable and unintended) change in a protocol-specific parameter or questionnaire response that is clinically relevant is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.


Status: Effective 

## 12.3 Procedures for Recording and Reporting AEs and SAEs

Subsequent to signing an ICF, all untoward medical occurrences that occur during the course of the study must be documented on the adverse event CRF. When possible, signs and symptoms indicating a common underlying pathology should be documented as one comprehensive event. For each recorded event, the AE documentation must include the onset date, outcome, resolution date (if event is resolved), intensity (ie, severity), any action with study treatment taken as a result of the event, and an assessment of the adverse event's relationship to the study treatment.

### **Nonserious Adverse Events**

A nonserious AE is defined as any untoward change in a subject's medical health that does not meet serious criteria noted below (eg, is not life-threatening, does not require hospitalization, does not prolong a current hospitalization, is not disabling, etc.). All adverse events must be reported regardless of whether or not they are related to the study treatment.

For nonserious adverse events, details should be entered on the adverse event CRF according to instructions provided by the Sponsor.

## **Serious Adverse Events**

A serious adverse event (SAE) is defined as any adverse experience that meets any of the following criteria:

- Results in death.
- Is life-threatening.

NOTE: Life-threatening means that the subject was at immediate risk of death from the reaction as it occurred, ie, it does not include a reaction which hypothetically might have caused death had it occurred in a more severe form

Requires inpatient hospitalization or prolongation of existing hospitalization.

NOTE: In general, hospitalization signifies that the individual remained at the hospital or emergency ward for observation and/or treatment (usually involving an overnight stay) that would not have been appropriate in the physician's office or an out-subject setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is


Status: Effective 

serious. When in doubt as to whether "hospitalization" occurred, the event should be considered serious.

 Results in persistent or significant disability/incapacity. Disability is defined as a substantial disruption of a person's ability to conduct normal life functions.

NOTE: The term disability means a substantial disruption of a person's ability to conduct normal life functions. This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, or accidental trauma (eg, sprained ankle) which may interfere or prevent everyday life functions but do not constitute a substantial disruption.

- Is a congenital anomaly/birth defect.
- Is an important medical event. An important medical event is an event that may not result in death, be life-threatening, or require hospitalization but may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in the definitions for SAEs. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in subject hospitalization, or the development of drug dependency or drug abuse.

All available information on a serious adverse event(s) and any other associated AE, if applicable, must be forwarded to the Sponsor immediately (ie, within 24 hours of the Investigator's or site's knowledge of the event) as follows:

- In studies utilizing EDC, all available information for the SAE and any associated AE(s) must be entered immediately into the EDC system.
  - Note: Should the EDC system become non-operational, the site must complete the appropriate Serious Adverse Event Form. The completed form is sent to the CTSO inbox email address: ct.suspected@novartis.com within 24 hours of the Investigator's or site's awareness; however, the reported information must be entered into the EDC system once it becomes operational.
- Sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.


Status: Effective 

 Additional information for any applicable event is to be reported as soon as it becomes available.

If the SAE is not previously documented in the Investigator's Brochure and is thought to be related to the investigational treatment the Sponsor may urgently require further information from the investigator for Health Authority reporting.

If the SAE was due to a hospitalization of the subject, a copy of the discharge summary should be made available to the Sponsor, upon request. In addition, a letter from the Investigator that summarizes the events related to the case as well as results of any relevant laboratory tests may also be requested. Further, depending upon the nature of the SAE, the Sponsor may request copies of applicable portions of the subject's medical records.

An assessment of seriousness will also be performed for all adverse events by a Sponsor physician utilizing the same criteria. If an adverse event reported for an Investigator's subject is upgraded to a serious adverse event by a Sponsor physician, the Investigator will receive a notification from the Sponsor.

In addition to the reporting of SAEs to the Sponsor, the SAE must be reported to the IEC / IRB according to their requirements.

Suspected Unexpected Serious Adverse Reactions (SUSARs) will be reported to the competent authorities and relevant ethics committees in accordance with EU Guidance 2011/C 172/01, or as per national regulatory requirements in participating countries. Sponsor may need to issue an Investigator Notification (IN) to inform all investigators involved in any study with the same investigational treatment that this SAE has been reported.

#### Adverse Events of Special Interest

An adverse event of special interest (ESI) is one of scientific and medical concern specific to the Sponsor's product or program where ongoing monitoring and rapid communication by the Investigator to the Sponsor may be appropriate. These adverse events may be serious or nonserious. Applicable adverse events may require further investigation in order to characterize and understand, and depending upon the nature of the event, rapid communication by the Sponsor to other parties may also be required.

The ESIs include the following:

Endophthalmitis


Status: Effective 

• Grade 3 aqueous flare and/or Grade 4 aqueous cells (see MOP for grading scale)

- Grade 2 aqueous flare and/or Grade 2 or 3 aqueous cells that fails to decrease to 1 or less within 30 days of the onset of the event (see MOP for grading scale)
- $\geq$  30 letter decrease in BCVA compared with Baseline visual acuity
- Sustained (> 15 minutes) loss of light perception due to elevated IOP
- IOP > 30 mmHg at/past 60 minutes postinjection
- Any elevation of IOP requiring surgical intervention (eg, paracentesis)
- New retinal tear or detachment
- New vitreous hemorrhage > 2+ severity that does not resolve within 14 days of the onset of the event (see MOP for grading scale)
- · New diagnosis of geographic atrophy
- Arterial thromboembolic events

## 12.4 Intensity and Causality Assessments

For every AE, the Investigator must assess the intensity (severity) and causality (relationship to study treatment). Specifically, AEs should be classified as mild, moderate, or severe. The assessment of causality will be based upon the categories of related and not related. These classifications should be based on the following definitions:

#### **Intensity (Severity):**

Mild An AE is mild if the subject is aware of, but can easily tolerate the sign

or symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort

significant enough to cause interference with the subject's usual

activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

**Causality:** 

Related An AE considered related to the use of the study treatment. AEs classified

as related may be either definitely related or possibly related where a

Print Date:


Status: Effective 

direct cause and effect relationship between the study treatment and the AE has not been demonstrated but there is a reasonable possibility that the AE was caused by the study treatment.

Not Related

An AE considered unrelated to the use of the study treatment. AEs classified as not related may either be definitely unrelated or simply unlikely to be related (ie, there are other more likely causes for the AE).

An assessment of causality will also be performed, when appropriate, by a Sponsor physician utilizing the same definitions. For a SAE reported by an Investigator as not related that is subsequently upgraded to be related by a Sponsor physician, the Investigator will receive a notification.

## 12.5 Unmasking of the Study Treatment

In case of emergency, information on the identity of the masked assigned IP is available to Investigators. If the treatment code needs to be broken in the interest of subject safety, the Investigator is encouraged to contact an appropriate unmasked Sponsor representative prior to unmasking if there is sufficient time. Dependent upon the individual circumstances (ie, medical emergency), the code may be broken by contacting the IRT system prior to contact with the Sponsor. The Sponsor must be informed in all cases in which the code was broken and of the circumstances involved.

Additionally, the Sponsor may be required to unmask the subject if the AE meets criteria of a SUSAR in order to fulfill expedited regulatory reporting requirements.

# 12.6 Follow-Up of Subjects with Adverse Events

The Investigator is responsible for adequate and safe medical care of subjects during the trial and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the trial. Any additional data from these follow-up procedures must be documented and available to the Sponsor.

# 12.7 Pregnancy in the Clinical Trial

Women of childbearing potential are not excluded from the study as long as adequate birth control methods are being utilized. Women of childbearing potential are defined as all women physiologically capable of becoming pregnant. Adequate birth control methods are summarized in the protocol's exclusion criteria.


Status: Effective 

Prior to enrollment in the study, female subjects of childbearing potential must be advised of the importance of avoiding pregnancy during the trial and the potential risks associated with an unintentional pregnancy. During the study, female subjects are to be instructed to contact the Investigator immediately if they suspect they might be pregnant. The Sponsor must be contacted immediately and a decision will be made regarding continuation of the pregnant woman in the study based upon the circumstances surrounding the pregnancy. Pregnancy is not reportable as an AE, however, complications may be reportable and will be decided on a case by case basis. A Sponsor prepared form will be utilized to capture all pregnancy-related information until birth of the child.

# 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

# 13.1 Completion of Source Documents and Electronic Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor. If electronic records are maintained, the method of verification must be determined in advance of starting the study. At a minimum, source documents should include the following information for each subject:

Subject identification (name, sex, race/ethnicity)

Documentation of subject eligibility

Date of informed consent

Dates of visits

Documentation that protocol specific procedures were performed

Results of study parameters, as required by the protocol

Study medication accountability records

Documentation of AEs and other safety parameters (if applicable)

Records regarding medical histories and the use of concomitant therapies prior to and during the study

Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.


Status: Effective 

Electronic case report forms will be provided to the sites; only designated individuals may complete the CRFs. The CRFs will be submitted at regular intervals based upon the study visit schedule. It is expected that all data reported will have corresponding entries in the source documents and that the Principal Investigator will review the reported data and certify that the CRFs are accurate and complete. No subject identifiers should be recorded on the CRFs beyond subject number and demographic information.

### 13.2 Data Review and Clarifications

The CRF data will be reviewed against the subject's source data by the study monitors to ensure completeness and accuracy. After monitoring has occurred at the clinical sites and the CRFs have been submitted, additional data clarifications and/or additions may be needed. Data clarifications and/or additions are documented and are part of each subject's CRFs.

## 13.3 Regulatory Documentation and Records Retention

The Investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the Sponsor, and the Investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is not subject to regulatory inspection and should be kept separately.

Additionally, the Investigator must keep study records and source documents until the Sponsor provides written approval for their destruction. If the Investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, the Sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations (generally 2 years after discontinuing clinical development or after the latest marketing approval).

# 13.4 Quality Assurance and Quality Control

The Sponsor will be responsible for implementing and maintaining quality assurance and quality control systems to ensure the study is conducted and data are generated, documented, and reported in compliance with the protocol, GCP and applicable regulatory requirements. The Sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the Sponsor, and inspection by domestic and foreign regulatory authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the Sponsor with the Investigator/Institution and any other parties involved in the study will be provided in writing as part of the protocol or as a separate agreement.


Status: Effective 

## 13.5 Data Monitoring Committee

An independent Data Monitoring Committee (DMC) will be established to monitor the safety of the trial participants, to ensure that the trial is being conducted with the highest scientific and ethical standards, and make appropriate recommendations based on the data seen.

The DMC charter will include the DMC membership and responsibilities, the timing of DMC meetings, the content of the analysis report for the DMC meetings, and the communications with the Sponsor. The DMC will only make recommendations for changes in study conduct.

### 14 REFERENCES

Bloch SB, Larsen M, Munch IC. Incidence of legal blindness from age-related macular degeneration in Denmark: Year 2000 to 2010. Am J Ophthalmol. 2012;153:209-13.

Brown DM, Kaiser PK, Michels M, Soubrane G, Heier JS, Kim RY, Sy JP et al. Ranibizumab versus verteporfin for neovascular age-related macular degeneration. N Engl J Med. 2009;355:1432-44.

Campbell JP, Bressler SB, Bressler NM. Impact of availability of anti-vascular endothelial growth factor therapy on visual impairment and blindness due to neovascular age-related macular degeneration. Arch Ophthalmol. 2012;130:794-5.

The CATT Research Group. Ranibizumab and Bevacizumab for Neovascular Age-Related Macular Degeneration. N Engl J Med. 2011;364:1897-1908.

Chong V, Amoaku W, Alsop J, Osborne A. Effectiveness of quarterly (Q3M) versus monthly (QM) ranibizumab according to initial gains in visual acuity - an analysis of 12 month data from the EXCITE study. 2013; 54:3816.

Ferris FL. Senile macular degeneration. Review of epidemiologic features. Am J Ophthalmol. 1983;118:132-51.

Ferris FL, Fine SL, Hyman L. Age-related macular degeneration and blindness due to neovascular maculopathy. Arch Ophthalmol. 1984;102:1640-42.

Heier JS, Brown DM, Chong V, Korobelnik JF, Kaiser PK, Nguyen QD et al. Intravitreal aflibercept (VEGF trap-eye) in wet age-related macular degeneration. Ophthalmology. 2012; 119:2537-48.


Status: Effective 

Kawasaki R, Yasuda M, Song S, Chen S-J, Jonas J, Wang J. The prevalence of age-related macular degeneration in Asians: A systematic review and meta-analysis. Ophthalmology. 2010;117:921-27.

Kim BJ, Ying GS, Huang J, Levy NE, Maguire MG, CATT Research Group. Sporadic visual acuity loss in the comparison of age-related macular degeneration treatments trials (CATT). Am J Ophthalmol. 2014;158:128-35.

Lim LS, Mitchell P, Seddon JM, Holz FG, Wong TY. Age-related macular degeneration. Lancet. 2012;379:1728-38.

Miller JW. Age-Related Macular Degeneration Revisited – Piecing the Puzzle: The LXIX Edward Jackson Memorial Lecture. Am J Ophthalmol. 2013;155:1-35.

Regillo CD, Brown DM, Abraham P, Yue H, Ianchulev T, Schneider S, Shams N. Randomized, double- masked, sham-controlled trial of ranibizumab for neovascular agerelated macular degeneration: PIER Study Year 1. Am J Ophthalmol 2008;145:239-48.

Rein DB, Wittenborn BS, Zhang X, Honeycutt AA, Lesesne SB, Saaddine J. Vision Health Cost-Effectiveness Study Group. Forecasting age-related macular degeneration through the year 2050. Arch Ophthalmol. 2009;127:533-40.

Rosenfeld PJ, Brown DM, Heier JS, Boyer DS, Kaiser PK, Chung CY et al. Ranibizumab for neovascular age-related macular degeneration. N Engl J Med. 2006;355:1419-31.

Schmidt-Erfurth U, Guymer Eldem B, Korobelnik JF, Schlingemann RO, Axer-Siegel R, Wiedemann P, et al. Efficacy and safety of monthly versus quarterly ranibizumab treatment in neovascular age-related macular degeneration: the EXCITE study. Ophthamology. 2011; 118: 831-39.

Schmidt-Erfurth U, Kaiser PK, Korobelnik JF, Brown DM, Chong V, Nguyen QD, et al. Intravitreal aflibercept injection for neovascular age-related macular degeneration: ninety-six-week results of the VIEW studies. Ophthalmology. 2014; 121:193-201.

Shah AR, Del Priore L V. Progressive visual loss in subfoveal exudation in age-related macular degeneration: a meta-analysis using Lineweaver-Burke plots. Am J Ophthalmol. 2007;143:83-89.

Shah AR, Del Priore LV. Natural history of predominantly classic, minimally classic and occult subgroups in age-related macular degeneration. Am J Ophthalmol. 2009;116:1901-07.


Status: Effective 

Simader C, Ritter M, Bolz M, Deak GG, Mayr-Sponer U, Golbaz I. Morphologic Parameters relevant for visual outcomes during anti-angiogenic therapy of neovascular age-related macular degeneration. Ophthalmology; 2014;121:1237-45.

Smith W, Assink J, Klein R, Mitchell P, Klaver CC, Klein BE. Risk factors for age-related macular degeneration: Pooled findings from three continents. Ophthalmology. 2001; 108:697-704.

Sommer A, Tielsch JM, Katz, J, Quigley HA, Gottsch JD, Javitt JC, Martone JF, Royall RM, Witt KA, Ezrine S. Racial differences in the cause-specific prevalence of blindness in East Baltimore. N Engl J Med. 1991;14:1412-17.

Spilsbury K, Garrett KL, Shen WY, Constable IJ, Rakoczy PE. Over expression of vascular endothelial growth factor (VEGF) in the retinal pigment epithelial leads to the development of choroidal neovascularization. Am J Pathol. 2000;157:135-44.

TAP and VIP Therapy Study Groups. Effect of lesion size, visual acuity and lesion composition on visual acuity change with and without verteporfin therapy for choroidal neovascularization secondary to age-related macular degeneration: TAP and VIP Report No.1. Am J Ophthalmol. 2003;136:407-18.

Wong TY, Chakravarthy U, Klein R, Mitchell P, Zlateva G, Buggage R, Fahrbach, K, Probst C, Sledge I. The natural history and prognosis of neovascular age-related macular degeneration: a systemic review of the literature and meta-analysis. Ophthalmology. 2008;115:116-26.

Ying GS, Kim BJ, Maguire MG, Huang J, Daniel E, Jaffe GJ, et al. Sustained visual acuity loss in the comparison of age-related macular degeneration treatments trials. JAMA Ophthalmol 2014:132:915-21.

### 15 APPENDIX

Not Applicable


Status: Effective